CLINICAL TRIAL: NCT02819635
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of Upadacitinib (ABT-494) for Induction and Maintenance Therapy in Subjects With Moderately to Severely Active Ulcerative Colitis
Brief Title: A Study to Evaluate the Safety and Efficacy of Upadacitinib (ABT-494) for Induction and Maintenance Therapy in Participants With Moderately to Severely Active Ulcerative Colitis (UC)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M14-234; 2016-000641-31 (EudraCT Number)
Record Dates: First submitted 2016-06-28; First posted 2016-06-30 (Estimated); Results first posted 2022-06-30 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Ulcerative Colitis (UC)
Keywords: Upadacitinib (ABT-494); Moderately to Severely Active UC; RINVOQ
MeSH Terms: conditions — Colitis, Ulcerative | interventions — upadacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (8):
- SS1: Placebo (Placebo Comparator): During the 8-week induction phase in Substudy 1, participants received placebo for upadacitinib film-coated tablets once daily by mouth (QD) for 8 weeks.
  Interventions: Drug: Placebo
- SS1: Upadacitinib 7.5 mg (Experimental): During the 8-week induction phase in Substudy 1, participants received 7.5 mg upadacitinib film-coated tablets once daily by mouth (QD) for 8 weeks.
  Interventions: Drug: Upadacitinib
- SS1: Upadacitinib 15 mg (Experimental): During the 8-week induction phase in Substudy 1, participants received 15 mg upadacitinib film-coated tablets once daily by mouth (QD) for 8 weeks.
  Interventions: Drug: Upadacitinib
- SS1: Upadacitinib 30 mg (Experimental): During the 8-week induction phase in Substudy 1, participants received 30 mg upadacitinib film-coated tablets once daily by mouth (QD) for 8 weeks. Additional participants were enrolled during the Substudy 1 analysis period and received 30 mg upadacitinib film-coated tablets once daily by mouth (QD) for 4 weeks.
  Interventions: Drug: Upadacitinib
- SS1: Upadacitinib 45 mg (Experimental): During the 8-week induction phase in Substudy 1, participants received 45 mg upadacitinib film-coated tablets once daily by mouth (QD) for 8 weeks. Additional participants were enrolled during the Substudy 1 analysis period and received 45 mg upadacitinib film-coated tablets once daily by mouth (QD) for 4 weeks.
  Interventions: Drug: Upadacitinib
- SS2: Placebo/Upadacitinib 45 mg (Experimental): During the Substudy 2 Part 1 induction period, participants received placebo for upadacitinib film-coated tablets once daily by mouth (QD) for 8 weeks. Participants who did not achieve clinical response at Week 8 of Part 1 were enrolled in an open-label extended treatment period and received 45 mg upadacitinib film-coated tablets once daily by mouth (QD) for an additional 8 weeks.
  Interventions: Drug: Placebo; Drug: Upadacitinib
- SS2: Upadacitinib 45 mg/Upadacitinib 45 mg (Experimental): During the Substudy 2 Part 1 induction period, participants received 45 mg upadacitinib film-coated tablets once daily by mouth (QD) for 8 weeks. Participants who did not achieve clinical response at Week 8 of Part 1 were enrolled in an open-label expended treatment period and received 45 mg upadacitinib film-coated tablets once daily by mouth (QD) for an additional 8 weeks.
  Interventions: Drug: Upadacitinib
- SS3: M14-675 clinical responders (Experimental): Participants in Study M14-675 (NCT03653026) who achieved clinical response defined by Adapted Mayo Score at Week 8 or Week 16 in that study and did not meet any study discontinuation criteria were eligible to enroll into Substudy 3. Participants were re-randomized and treated with a blinded treatment assignment (15 mg upadacitinib film-coated tablets once daily by mouth [QD], or 30 mg upadacitinib film-coated tablets QD, or placebo for upadacitinib film-coated tablets QD) for up to 52 weeks.
  Interventions: Drug: Placebo; Drug: Upadacitinib

INTERVENTIONS:
Drug: Placebo — Film-coated tablet for oral administration
  Arms: SS1: Placebo; SS2: Placebo/Upadacitinib 45 mg; SS3: M14-675 clinical responders
Drug: Upadacitinib — Film-coated tablet for oral administration
  Other Names: ABT-494; RINVOQ
  Arms: SS1: Upadacitinib 15 mg; SS1: Upadacitinib 30 mg; SS1: Upadacitinib 45 mg; SS1: Upadacitinib 7.5 mg; SS2: Placebo/Upadacitinib 45 mg; SS2: Upadacitinib 45 mg/Upadacitinib 45 mg; SS3: M14-675 clinical responders

SUMMARY:
This study was comprised of three substudies. The objective of Substudy 1 was to characterize the dose-response, efficacy, and safety of upadacitinib compared to placebo in inducing clinical remission to identify the induction dose of upadacitinib for further evaluation in Substudy 2. The objective of Substudy 2 was to evaluate the efficacy and safety of upadacitinib compared to placebo in inducing clinical remission in participants. The objective of Substudy 3 was to evaluate the efficacy and safety of upadacitinib compared to placebo in achieving clinical remission in participants who had a response following induction with upadacitinib.

DETAILED DESCRIPTION:
Substudy 1 was a Phase 2b dose-ranging study designed to evaluate the efficacy and safety of different oral doses of upadacitinib compared to placebo as 8-week induction therapy in participants with moderately to severely active UC. Approximately 250 participants were planned to be randomized 1:1:1:1:1 to the placebo group and 4 upadacitinib doses (7.5, 15, 30, and 45 mg). Randomization was stratified by previous biologic therapy use (yes/no), Baseline corticosteroid use (yes/no), and Baseline Adapted Mayo score (≤ 7 or > 7). The study duration included a Screening Period of up to 5 weeks and an 8-week double-blind (DB) Induction Period. After all randomized participants completed the 8-week induction, a dose-selection analysis of efficacy and safety (selected laboratory parameters) of upadacitinib versus placebo was performed. Based on this dose-selection analysis, one induction dose (upadacitinib 45 mg) was identified for further evaluation in two Phase 3 induction studies, M14-234 Substudy 2 and M14-675 (NCT03653026). During the analysis period, 132 additional participants were randomized into Groups 3 and 4 of Substudy 1 (upadacitinib 30 mg and 45 mg dose groups; approximately 66 participants per dose group). The objectives of enrolling these additional participants were to avoid interrupting the study activities during the analysis period and to support a sufficient number of participants with clinical response to be re-randomized into the maintenance portion in Substudy 3. Substudy 1 main participants are defined as those first 250 randomized 250, and additional participants are defined as those who were randomized after the main participants.

Substudy 2 was a two-part Phase 3 dose-confirming study designed to evaluate the efficacy and safety of oral administration of upadacitinib 45 mg compared to placebo as induction therapy for up to 16 weeks in participants with moderately to severely active UC. Substudy 2 included a Screening Period of up to 5 weeks, Part 1, and Part 2. Part 1 was a randomized, DB, placebo-controlled 8-week induction period. Part 2 was an open-label, 8-week extended treatment period for clinical non-responders from Part 1 of Substudy 2. Part 1 was planned to enroll 462 subjects; actual enrollment was 474 subjects. Eligible participants were randomized in a 2:1 ratio to one of the two treatment groups (DB upadacitinib 45 mg or matching placebo) for 8 weeks. The randomization was stratified by bio-IR status (Biologic inadequate responders [bio-IR] vs Non-biologic-inadequate responders [non-bio-IR], corticosteroid use (yes or no), and Adapted Mayo score (≤ 7 or > 7) at Baseline. Within bio-IR, the randomization was further stratified by number of prior biologic treatments (≤ 1 or > 1). Within non-bio-IR, the randomization was further stratified by previous biologic use (yes or no). Part 2 was an open label, 8-week Extended Treatment Period for those who did not achieve clinical response per Adapted Mayo score at Week 8 in Part 1. All participants received upadacitinib 45 mg.

Substudy 3 was a Phase 3 maintenance study designed to evaluate the efficacy and safety of upadacitinib 15 and 30 mg once daily (QD) compared to placebo in achieving clinical remission per Adapted Mayo score in participants with moderately to severely active UC who achieved clinical response per Adapted Mayo score following induction therapy from Substudy 1, Substudy 2, or Study M14-675. A total of 1,046 subjects who achieved clinical response per Adapted Mayo score after completion of induction treatment or Extended Treatment Period in Study M14-234 Substudy 1, Substudy 2, or Study M14-675 entered Substudy 3, and 1,044 were treated with a blinded treatment assignment for up to 52 weeks. Substudy 3 included 4 cohorts. Cohort 1: 847 participants who achieved clinical response in Substudy 1, Substudy 2, or Study M14-675 at either Week 8 or Week 16, and received upadacitinib 15, 30, or 45 mg QD. The treatment groups in Cohort 1 were Group 1: upadacitinib 15 mg QD; Group 2: upadacitinib 30 mg QD; and Group 3: placebo QD. Those who achieved clinical response and received upadacitinib 15 mg QD in Substudy 1 were re-randomized 1:1 to only receive upadacitinib 15 mg QD or placebo QD (treatment Group 1 or 3). Cohort 2: 104 participants who received double-blind placebo QD treatment for 8 weeks during Substudy 1, Substudy 2 Part 1, or Study M14-675 Part 1 and achieved clinical response at Week 8 continued to receive blinded placebo QD in Substudy 3. Cohort 3: 75 participants who received upadacitinib 45 mg QD in Induction Phase and did not achieve clinical response and received upadacitinib 45 mg QD in Extended Treatment in Substudy 2 Part 2 or in Study M14-675 Part 2 and achieved clinical response at Week 16 were re-randomized 1:1 and received blinded upadacitinib 30 mg QD or upadacitinib 15 mg QD in Substudy 3. Cohort 4: 20 participants who received double-blinded treatment of upadacitinib 7.5 mg QD for 8 weeks during Substudy 1 and achieved clinical response at Week 8 continued to receive blinded treatment of upadacitinib 7.5 mg QD in Substudy 3.

ELIGIBILITY:
Inclusion Criteria:

Note: Adolescent participants who are 16 or 17 years old will be eligible to participate if approved by the country or regulatory/health authority. If approval has not been granted, only participants ≥18 years old will be enrolled. Adolescents must weigh ≥ 40 kilograms and meet the definition of Tanner Stage 5 at Screening Visit.

* Diagnosis of ulcerative colitis for 90 days or greater prior to Baseline, confirmed by colonoscopy during the Screening Period, with exclusion of current infection, colonic dysplasia and/or malignancy. Appropriate documentation of biopsy results consistent with the diagnosis of UC, in the assessment of the Investigator, must be available.
* Active ulcerative colitis with an Adapted Mayo score of 5 to 9 points and endoscopic sub score of 2 to 3 (confirmed by central reader).
* Demonstrated an inadequate response to, loss of response to, or intolerance to at least one of the following treatments including: oral aminosalicylates, corticosteroids, immunosuppressants, and/or biologic therapies in the opinion of the investigator.

Note: Participants who have had inadequate response, loss of response to conventional therapy, but have not failed biologic therapy (Non-bio-IR) and have received a prior biologic for up to 1 year may be enrolled, however they must have discontinued the biologic for reasons other than inadequate response or intolerance (e.g., change of insurance, well controlled disease) and must meet criteria for inadequate response, loss of response or intolerance to aminosalicylates, corticosteroids, and/or immunosuppressants as defined above.

* If female, participant must meet the criteria for Contraception Recommendations
* Female participants of childbearing potential must have a negative serum pregnancy test at the Screening Visit and a negative urine pregnancy test at the Baseline Visit prior to study drug dosing.

Exclusion Criteria:

* Participant with current diagnosis of Crohn's disease (CD) or diagnosis of indeterminate colitis (IC)
* Current diagnosis of fulminant colitis and/or toxic megacolon
* Participant with disease limited to the rectum (ulcerative proctitis) during the screening endoscopy
* Received cyclosporine, tacrolimus, mycophenolate mofetil, or thalidomide within 30 days prior to Baseline
* Participant on azathioprine or 6-mercaptopurine within 10 days of Baseline
* Received intravenous corticosteroids within 14 days prior to Screening or during the Screening Period.
* Participant with previous exposure to Janus Activated Kinase (JAK) inhibitor (e.g., tofacitinib, baricitinib, filgotinib, upadacitinib).
* Screening laboratory and other analyses show any abnormal results meeting the exclusion criteria

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1302 (Actual)
Dates: Start 2016-09-26 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2021-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (496):
- United States (149):
  - Birmingham Gastroenterology Associates P.C /ID# 151276, Birmingham, Alabama
  - East View Medical Research, LLC /ID# 171183, Mobile, Alabama
  - CB Flock Research Corporation /ID# 165980, Mobile, Alabama
  - Delsol Research Management, Ll /Id# 170131, Chandler, Arizona
  - Digestive Disease Consultants, A Division of Arizona Digestive Health, P.C /ID# 211885, Mesa, Arizona
  - Arizona Arthritis & Rheumatology Research, PLLC /ID# 169822, Sun City, Arizona
  - Adobe Clinical Research LLC /ID# 155250, Tucson, Arizona
  - University of Arizona /ID# 150553, Tucson, Arizona
  - Citrus Valley Gastroenterology /ID# 151914, Covina, California
  - Newport Huntington Medical Group /ID# 217005, Huntington Beach, California
  - UC San Diego Health System /ID# 155185, La Jolla, California
  - United Medical Doctors /ID# 207464, Los Alamitos, California
  - TLC Clinical Research Inc /ID# 216829, Los Angeles, California
  - Gastrointestinal Biosciences Clinical Trials, LLC /ID# 157080, Los Angeles, California
  - Facey Medical Foundation /ID# 203133, Mission Hills, California
  - United Medical Doctors - Murrieta /ID# 151211, Murrieta, California
  - InSite Digestive Health Care - Oxnard /ID# 163414, Oxnard, California
  - Inland Empire Clinical Trials, LLC /ID# 216038, Rialto, California
  - San Diego Clinical Trials /ID# 212120, San Diego, California
  - Medical Assoc Research Grp /ID# 169148, San Diego, California
  - Univ of California San Francis /ID# 164581, San Francisco, California
  - Delta Waves, Inc. /ID# 151721, Colorado Springs, Colorado
  - South Denver Gastroenterology /ID# 151223, Lone Tree, Colorado
  - Western States Clinical Res /ID# 158076, Wheat Ridge, Colorado
  - Western Connecticut Medical Group /ID# 169210, Danbury, Connecticut
  - Medical Research Center of CT /ID# 150482, Hamden, Connecticut
  - Gastro Florida /ID# 155245, Clearwater, Florida
  - Moonshine Research Center, Inc /ID# 152533, Doral, Florida
  - Universal Axon Clinical Research /ID# 213461, Doral, Florida
  - Palmetto Research, LLC /ID# 151716, Hialeah, Florida
  - Nature Coast Clinical Research - Inverness /ID# 154064, Inverness, Florida
  - Encore Borland-Groover Clinical Research /Id# 170912, Jacksonville, Florida
  - SIH Research Mumtaz, Inc /ID# 163319, Kissimmee, Florida
  - Cfagi Llc /Id# 202017, Maitland, Florida
  - University of Miami /ID# 215441, Miami, Florida
  - Advanced Pharma /ID# 151719, Miami, Florida
  - New Horizon Research Center /ID# 152474, Miami, Florida
  - Crystal Pharmacology Research /ID# 151841, Miami, Florida
  - Coral Research Clinic /ID# 150444, Miami, Florida
  - Advanced Research Institute, Inc /ID# 163098, New Port Richey, Florida
  - Endoscopic Research, Inc. /ID# 151720, Orlando, Florida
  - Omega Research Maitland, LLC /ID# 200269, Orlando, Florida
  - Clinical Research Trials of Florida, Inc. /ID# 201790, Tampa, Florida
  - University of South Florida /ID# 214493, Tampa, Florida
  - AdventHealth Tampa /ID# 200272, Tampa, Florida
  - Gastroenterology Associates of Central Georgia, LLC /ID# 165782, Macon, Georgia
  - Infinite Clinical Trials /ID# 215340, Riverdale, Georgia
  - Atlanta Gastroenterology Spec /ID# 150548, Suwanee, Georgia
  - Next Innovative Clinical Research - Chicago /ID# 216060, Chicago, Illinois
  - The University of Chicago DCAM /ID# 150547, Chicago, Illinois
  - NorthShore University HealthSystem /ID# 150555, Evanston, Illinois
  - Northwest Health Care Associates /ID# 151590, Hoffman Estates, Illinois
  - Carle Foundation Hospital /ID# 151137, Urbana, Illinois
  - MediSphere Medical Research Center /ID# 152064, Evansville, Indiana
  - Indianapolis Gastroenterology /ID# 162901, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics /ID# 157058, Iowa City, Iowa
  - Cotton-O'Neil Clinical Res Ctr /ID# 167182, Topeka, Kansas
  - Tri-State Gastroenterology /ID# 169811, Crestview Hills, Kentucky
  - Houma Digestive Health Special /ID# 151844, Houma, Louisiana
  - Nola Research Works, LLC /ID# 153356, New Orleans, Louisiana
  - Louisana Research Center, LLC /ID# 150446, Shreveport, Louisiana
  - University of Maryland Med Ctr /ID# 150449, Baltimore, Maryland
  - Gastro Center of Maryland /ID# 200022, Columbia, Maryland
  - Massachusetts General Hospital /ID# 165676, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center Michigan Medicine /ID# 151140, Ann Arbor, Michigan
  - Huron Gastroenterology Assoc /ID# 152710, Ann Arbor, Michigan
  - Clin Res Inst of Michigan, LLC /ID# 153027, Chesterfield, Michigan
  - Revival Research Institute, LLC /ID# 207280, Southfield, Michigan
  - Center for Digestive Health /ID# 161984, Troy, Michigan
  - Gastroenterology Associates of Western Michigan, PLC d.b.a. West Michigan Clinic /ID# 157484, Wyoming, Michigan
  - Mayo Clinic - Rochester /ID# 151677, Rochester, Minnesota
  - Minnesota Gastroenterology PA /ID# 151678, Saint Paul, Minnesota
  - University of Mississippi Medical Center /ID# 213139, Jackson, Mississippi
  - Southern Therapy and Advanced Research (STAR) LLC /ID# 170712, Jackson, Mississippi
  - Washington University-School of Medicine /ID# 150485, St Louis, Missouri
  - Las Vegas Medical Research /ID# 153044, Las Vegas, Nevada
  - Dartmouth-Hitchcock Medical Center /ID# 150549, Lebanon, New Hampshire
  - AGA Clinical Research Associates, LLC /ID# 153040, Egg Harbor, New Jersey
  - Atlantic Digestive Health Inst /ID# 150447, Morristown, New Jersey
  - Rutgers Robert Wood Johnson /ID# 155248, New Brunswick, New Jersey
  - Duplicate_University of New Mexico Department of Internal Medicine /ID# 214396, Albuquerque, New Mexico
  - NY Scientific /ID# 152707, Brooklyn, New York
  - NYU Langone Long Island Clinical Research Association /ID# 155272, Great Neck, New York
  - Columbia Univ Medical Center /ID# 163410, New York, New York
  - DiGiovanna Institute for Medical Education & Research /ID# 201533, North Massapequa, New York
  - Premier Medical Group - GI Division /ID# 153357, Poughkeepsie, New York
  - Gastoenterology Group of Rochester /ID# 151079, Rochester, New York
  - Richmond University Medical Center /ID# 201859, Staten Island, New York
  - Montefiore Medical Center - Moses Campus /ID# 150543, The Bronx, New York
  - Advantage Clinical Trials /ID# 163938, The Bronx, New York
  - Digestive Health Partners, P.A /ID# 167237, Asheville, North Carolina
  - Atrium Health Carolinas Medical Center /ID# 156971, Charlotte, North Carolina
  - Charlotte Gastroenterology and Hepatology, PLLC /ID# 150545, Charlotte, North Carolina
  - Atlantic Gastroenterology Clinical Research /ID# 151899, Greenville, North Carolina
  - Clinical Trials of America /ID# 153448, Winston-Salem, North Carolina
  - Wake Forest Baptist Medical Center /ID# 150448, Winston-Salem, North Carolina
  - Plains Clinical Research Center, LLC /ID# 170290, Fargo, North Dakota
  - Consultants for Clinical Research /ID# 151679, Cincinnati, Ohio
  - University of Cincinnati /ID# 164582, Cincinnati, Ohio
  - The Ohio State University /ID# 169416, Columbus, Ohio
  - Optimed Research, Ltd. /ID# 169696, Columbus, Ohio
  - Hometown Urgent Care and Resea /ID# 200065, Dayton, Ohio
  - Dayton Gastroenterology, Inc. /ID# 167631, Englewood, Ohio
  - Great Lakes Medical Research, LLC /ID# 201772, Mentor, Ohio
  - Ohio Clinical Research Partner /ID# 154068, Mentor, Ohio
  - Hightower Clinical /ID# 216337, Oklahoma City, Oklahoma
  - Digestive Disease Specialists /ID# 201056, Oklahoma City, Oklahoma
  - Options Health Research, LLC /ID# 150554, Tulsa, Oklahoma
  - Healthcare Research Consultant /ID# 163100, Tulsa, Oklahoma
  - Northwest Gastroenterology Clinic /ID# 152527, Portland, Oregon
  - Guthrie Medical Group, PC /ID# 150481, Sayre, Pennsylvania
  - Penn State Health Colonnade /ID# 150259, State College, Pennsylvania
  - Pharmacorp Clinical Trials /ID# 153354, Charleston, South Carolina
  - Gastroenterology Associates, P.A. of Greenville /ID# 150541, Greenville, South Carolina
  - Gastro One /ID# 151144, Germantown, Tennessee
  - East Tennessee Research Institute /ID# 203610, Johnson City, Tennessee
  - Quality Medical Research /ID# 203426, Nashville, Tennessee
  - Vanderbilt University Medical Center /ID# 153355, Nashville, Tennessee
  - TX Clinical Research Institute /ID# 151526, Arlington, Texas
  - Inquest Clinical Research /ID# 164635, Baytown, Texas
  - Texas Digestive Disease Consultants /ID# 209947, Cedar Park, Texas
  - Texas Digestive Disease Consultants /ID# 209804, Cedar Park, Texas
  - Baylor Scott & White Center for Inflammatory Bowel Diseases /ID# 200770, Dallas, Texas
  - DHAT Research Institute /ID# 151218, Garland, Texas
  - Vilo Research Group Inc /ID# 212624, Houston, Texas
  - CliniCore International, LLC /ID# 152062, Houston, Texas
  - Baylor College of Medicine - Baylor Medical Center /ID# 150486, Houston, Texas
  - Centex Studies, Inc. - Houston /ID# 201216, Houston, Texas
  - GI Specialists of Houston /ID# 202327, Houston, Texas
  - Caprock Gastro Research, LLC /ID# 214754, Lubbock, Texas
  - Clinical Associates in Research Therapeutics of America, LLC /ID# 201260, San Antonio, Texas
  - Southern Star Research Institute, LLC /ID# 169396, San Antonio, Texas
  - Carl R. Meisner Medical Clinic /ID# 171061, Sugar Land, Texas
  - Baylor Scott & White Center for Diagnostic Medicine /ID# 204499, Temple, Texas
  - Tyler Research Institute, LLC /ID# 169146, Tyler, Texas
  - Gastro Health & Nutrition - Victoria /ID# 167761, Victoria, Texas
  - HP Clinical Research /ID# 163939, Bountiful, Utah
  - Advanced Research Institute /ID# 162624, Ogden, Utah
  - Utah Gastroenternology - St. Mark's Office /ID# 163101, Salt Lake City, Utah
  - Velocity Clinical Research - Salt Lake City /ID# 163181, West Jordan, Utah
  - Ctr for Gastrointestinal Healt /ID# 153360, Franklin, Virginia
  - Emeritas Research Group, LLC /ID# 150258, Leesburg, Virginia
  - Washington Gastroenterology /ID# 163629, Bellevue, Washington
  - Virginia Mason Medical Center /ID# 153026, Seattle, Washington
  - The Polyclinic /ID# 164369, Seattle, Washington
  - The Vancouver Clinic, INC. PS /ID# 162333, Vancouver, Washington
  - Aurora Medical Center - Grafto /ID# 151717, Grafton, Wisconsin
  - Wisconsin Center for Advanced Research, a division of GI Associates, LLC /ID# 151838, Milwaukee, Wisconsin
  - Medical College of Wisconsin /ID# 151843, Milwaukee, Wisconsin
- Argentina (6):
  - Cardio Alem /ID# 211280, San Isidro, Buenos Aires
  - Gedyt /ID# 210015, Ciudad Autonoma de Buenos Aire, Ciuadad Autonoma de Buenos Aires
  - Mautalen Salud e Investigacion /ID# 171173, Ciudad Autonoma de Buenos Aire, Ciuadad Autonoma de Buenos Aires
  - Hospital Britanico de Buenos Aires /ID# 209495, Ciudad Autonoma de Buenos Aire, Ciuadad Autonoma de Buenos Aires
  - Sanatorio 9 de Julio /ID# 150189, San Miguel de Tucumán, Tucumán Province
  - Hospital Privado Univesitario /ID# 164185, Córdoba
- Australia (6):
  - Macquarie University Hospital /ID# 211951, Macquarie University, New South Wales
  - Mater Misericordiae Limited /ID# 212685, South Brisbane, Queensland
  - Griffith University /ID# 211952, Southport, Queensland
  - Monash Medical Centre /ID# 150206, Clayton, Victoria
  - St Vincent's Hospital Melbourne /ID# 152472, Fitzroy Melbourne, Victoria
  - Fiona Stanley Hospital /ID# 211640, Murdoch, Western Australia
- Austria (4):
  - Ordensklinikum Linz GmbH Barmherzige Schwestern /ID# 150305, Linz, Upper Austria
  - Klinik Landstrasse /ID# 162866, Vienna, Vienna
  - Medizinische Universitaet Wien /ID# 150614, Vienna, Vienna
  - Landeskrankenhaus Salzburg-Universitätsklinikum der PMU (LKH) /ID# 150306, Salzburg
- Vitebsk Regional Advanced Clin /ID# 169612, Vitebsk, Belarus
- Belgium (3):
  - Universitair Ziekenhuis Leuven /ID# 150332, Leuven, Vlaams-Brabant
  - AZ Maria Middelares /ID# 150331, Ghent
  - AZ-Delta /ID# 150330, Roeselare
- Bosnia and Herzegovina (5):
  - University Clinical Centre of the Republic of Srpska /ID# 150209, Banja Luka, Republika Srpska
  - University Clinical Centre of the Republic of Srpska /ID# 150706, Banja Luka, Republika Srpska
  - University Clinical Center Tuzla /ID# 150211, Tuzla, Tuzlanski
  - University Clinical Hospital Mostar /ID# 150705, Mostar
  - Clinical Center University of Sarajevo /ID# 150208, Sarajevo
- Brazil (7):
  - Instituto Goiano de Gastroenterologia e Endoscopia Digestiva /ID# 153742, Goiânia, Goiás
  - Hospital Nossa Senhora das Graças /ID# 152480, Curitiba, Paraná
  - Hospital de Clinicas de Porto Alegre /ID# 153743, Porto Alegre, Rio Grande do Sul
  - Upeclin Fmb - Unesp /Id# 152485, Botucatu, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina de Ribeirao Preto - USP /ID# 152484, Ribeirão Preto, São Paulo
  - Faculdade de Medicina do ABC /ID# 152481, Santo André, São Paulo
  - Kaiser Clinica e Hospital Dia /ID# 152483, São José do Rio Preto, São Paulo
- Canada (16):
  - University of Calgary /ID# 151821, Calgary, Alberta
  - Allen Whey Khye Lim Professional Corporation /ID# 211168, Edmonton, Alberta
  - University of Alberta - Zeidler Ledcor Centre /ID# 151100, Edmonton, Alberta
  - Covenant Health /ID# 158930, Edmonton, Alberta
  - Okanagan Clinical Trials /ID# 153178, Kelowna, British Columbia
  - Percuro Clinical Research, Ltd /ID# 150367, Victoria, British Columbia
  - Medicor Research Inc /ID# 151101, Greater Sudbury, Ontario
  - Hamilton Health Sciences - McMaster University Medical Centre /ID# 150365, Hamilton, Ontario
  - Ottawa Hospital Research Institute /ID# 151820, Ottawa, Ontario
  - Toronto Digestive Disease Asso /ID# 150363, Vaughan, Ontario
  - CISSS de la Monteregie /ID# 159215, Greenfield Park, Quebec
  - CISSS de Chaudière-Appalaches, Hôpital Hotel-Dieu de Lévis /ID# 150361, Lévis, Quebec
  - Recherche GCP Research /ID# 151822, Montreal, Quebec
  - Centre Hospitalier de l'Universite de Montreal - CRCHUM /ID# 167169, Montreal, Quebec
  - Montreal General Hospital - McGill University Health Centre /ID# 170012, Montreal, Quebec
  - CIUSSS de l'Estrie - CHUS /ID# 150366, Sherbrooke, Quebec
- Chile (6):
  - M y F Estudios Clínicos /ID# 200107, Santiago, Region Metropolitana Santiago
  - Centro de Investigaciones Clínicas Viña del Mar /ID# 150212, Viña del Mar, Región de Valparaíso
  - Research Group /ID# 203176, Santiago, Santiago Metropolitan
  - Hospital Guillermo Grant Benavente de Concepción /ID# 212424, Concepción
  - CTR Estudios Clinicos /ID# 200110, Providencia
  - Hospital Clinico Universidad De Los Andes /ID# 207422, Santiago
- China (16):
  - The First Affiliated Hospital, Sun Yat-sen University /ID# 150455, Guangzhou, Guangdong
  - The Sixth Affiliated Hosp Sun /ID# 150456, Guangzhou, Guangdong
  - Affiliated Taihe Hospital of Hubei University of Medicine /ID# 216405, Shiyan, Hubei
  - Tongji Hospital Tongji Medical College Huazhong University of Science and Techno /ID# 167088, Wuhan, Hubei
  - Union Hospital Tongji Medical College Huazhong University of Science and Technol /ID# 167078, Wuhan, Hubei
  - The First Affiliated Hospital of Nanchang University /ID# 211750, Nanchang, Jiangxi
  - The First Hospital of Jilin University /ID# 209986, Changchun, Jilin
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine /ID# 150461, Shanghai, Shanghai Municipality
  - Shanghai Tenth People's Hospital /ID# 150460, Shanghai, Shanghai Municipality
  - Renji Hospital, Shanghai Jiaotong University School of Medicine /ID# 165815, Shanghai, Shanghai Municipality
  - The second Affiliated hospital of Zhejiang University school of Medicine /ID# 165807, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital,Meical School Zhejiang University /ID# 150454, Hangzhou, Zhejiang
  - Xiangya Hospital Central South University /ID# 167229, Changsha
  - West China Hospital, Sichuan University /ID# 167040, Chengdu
  - Shengjing Hospital of China Medical University /ID# 166920, Shenyang
  - Tianjin Medical University General Hospital /ID# 170604, Tianjin
- Colombia (3):
  - Corporacion Hospitalaria Juan Cuidad Sede Denominada Hospital Universitario Mayo /ID# 151564, Bogota DC, Cundinamarca
  - Instituto Medico de Alta Tecnologia Oncomédica S.A /ID# 207042, Montería, Departamento de Córdoba
  - Hospital Universitario de San /ID# 155387, Medellín
- Croatia (8):
  - Clinical Hospital Dubrava /ID# 150213, Zagreb, City of Zagreb
  - Klinicki bolnicki centar Zagreb /ID# 150225, Zagreb, City of Zagreb
  - Klinicki bolnicki centar Zagreb /ID# 150709, Zagreb, City of Zagreb
  - Poliklinika Solmed /ID# 211483, Zagreb, City of Zagreb
  - Duplicate_Klinicki bolnicki centar Osijek /ID# 150216, Osijek, County of Osijek-Baranja
  - Klinicki bolnicki centar Rijeka /ID# 150708, Rijeka, Primorje-Gorski Kotar County
  - Klinicki bolnicki centar Split /ID# 213988, Split, Split-Dalmatia County
  - Zadar General Hospital /ID# 150221, Zadar
- Czechia (7):
  - Hepato-Gastroenterologie HK, s.r.o. /ID# 150912, Hradec Králové
  - CTCenter MaVe s.r.o. /ID# 150904, Olomouc
  - ARTROSCAN s.r.o. /ID# 150401, Ostrava
  - Nemocnice Pardubickeho kraje, a.s. /ID# 213539, Pardubice
  - Nemocnice Milosrdnych sester sv. Karla Boromejskeho v Praze /ID# 216221, Prague
  - Axon Clinical, s.r.o. /ID# 152479, Prague
  - ISCARE a.s. /ID# 209278, Prague
- Estonia (4):
  - East Tallinn Central Hospital /ID# 150417, Kesklinn, Harju
  - North Estonia Medical Centre /ID# 160870, Mustamäe, Harju
  - Tartu University Hospital /ID# 150418, Tartu, Tartu
  - West Tallinn Central Hospital /ID# 150419, Tallinn
- Finland (5):
  - Tampere University Hospital /ID# 150114, Tampere, Pirkanmaa
  - Duplicate_Helsinki Univ Central Hospital /ID# 150407, Helsinki
  - Keski-Suomen Sairaala Nova /ID# 155666, Jyväskylä
  - Laakarikeskus Ikioma /ID# 150121, Mikkeli
  - Turku University Hospital /ID# 168301, Turku
- France (8):
  - Chu de Nice-Hopital L'Archet Ii /Id# 152606, Nice, Alpes-Maritimes
  - HCL - Hôpital Lyon Sud /ID# 152539, Pierre-Bénite, Auvergne-Rhône-Alpes
  - CHU Hopital Nord /ID# 163508, Marseille, Bouches-du-Rhone
  - CHRU Lille - Hopital Claude Huriez /ID# 152607, Lille, Hauts-de-France
  - CHU Montpellier - Hôpital Saint Eloi /ID# 200006, Montpellier, Herault
  - CHU Amiens-Picardie Site Sud /ID# 163456, Amiens, Somme
  - CHD Vendée- La Roche-sur-Yon - Les Oudairies /ID# 154452, La Roche-sur-Yon
  - CHU de Saint-Etienne, Hopital Nord /ID# 154453, Saint-Etienne
- Germany (10):
  - Universitatsklinikum Mannheim /ID# 150173, Mannheim, Baden-Wurttemberg
  - Universitaetsklinimum Tuebingen /ID# 150767, Tübingen, Baden-Wurttemberg
  - Universitatsklinikum Munster /ID# 150158, Munster, Lower Saxony
  - Gastroenterologische Gemeinschaftspraxis Herne /ID# 214574, Herne, North Rhine-Westphalia
  - Zentrum für Gastroenterologie Saar MVZ GmbH /ID# 215811, Saarbrücken, Saarland
  - Universitaetsklinikum Schleswig-Holstein Campus Kiel /ID# 161981, Kiel, Schleswig-Holstein
  - MVZ fuer Gastroenterlogie am Bayerischen Platz /ID# 150766, Berlin
  - Agaplesion Markus Krankenhaus /ID# 161982, Frankfurt am Main
  - Medizinisches Versorgungszentrum Portal 10 /ID# 207135, Münster
  - Praxis medicum /ID# 150166, Wiesbaden
- Greece (7):
  - General Hospital of Athens Laiko /ID# 208669, Athens, Attica
  - General Hospital of Chest Diseases of Athens SOTIRIA /ID# 202100, Athens, Attica
  - University General Hospital of Heraklion PA.G.N.I /ID# 150250, Heraklion, Crete
  - General Hospital of Athens Evaggelismos and Ophthalmiatrio of Athens Polyclinic /ID# 150309, Athens
  - University General Hospital of Ioannina /ID# 164248, Ioannina
  - Theageneio Anticancer Hospital /ID# 163896, Thessaloniki
  - General Hospital of Thessaloniki Hippokrateio /ID# 209521, Thessaloniki
- Hungary (6):
  - Markusovszky Egyetemi Oktatokorhaz /ID# 150313, Szombathely, Vas County
  - Bekes Megyei Kozponti Korhaz /ID# 151572, Békéscsaba
  - Semmelweis Egyetem /ID# 150312, Budapest
  - Meditres Kft. /ID# 151521, Kecskemét
  - Soproni Erzsebet Oktato Korhaz es Rehabilitacios Intezet /ID# 151523, Sopron
  - Mentahaz Maganorvosi Kozpont /ID# 205884, Székesfehérvár
- Ireland (5):
  - Beaumont Hospital /ID# 150321, Beaumont, Dublin
  - St James Hospital /ID# 150320, Dublin, Dublin
  - St Vincent's University Hospital /ID# 150318, Elm Park, Dublin
  - Mercy University Hospital /ID# 151529, Cork
  - University Hospital Galway /ID# 150319, Galway
- Israel (4):
  - Soroka University Medical Center /ID# 156561, Beersheba, Southern District
  - Rambam Health Care Campus /ID# 150325, Haifa
  - Shaare Zedek Medical Center /ID# 161677, Jerusalem
  - Hadassah Medical Center-Hebrew University /ID# 165118, Jerusalem
- Italy (10):
  - Azienda Ospedaliera San Camillo Forlanini /ID# 151360, Rome, Lazio
  - ASST Rhodense/Presidio Ospedaliero di Rho /ID# 216610, Rho, Milano
  - Istituto Clinico Humanitas /ID# 151361, Rozzano, Milano
  - Fondazione PTV Policlinico Tor Vergata /ID# 150338, Rome, Roma
  - Presidio Columbus-Fondazione Policlinico Universitario Agostino Gemelli IRCCS-Un /ID# 150333, Rome, Roma
  - IRCCS Ospedale Sacro Cuore Don Calabria /ID# 201725, Negrar, Verona
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna /ID# 150337, Bologna
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico /ID# 150334, Milan
  - ASST Fatebenefratelli Sacco - Ospedale Fatebenefratelli e Oftalmico /ID# 150602, Milan
  - A.O. Ospedali Riuniti Villa Sofia - Cervello /ID# 150253, Palermo
- Japan (73):
  - Aichi Medical University Hospital /ID# 151993, Nagakute-shi, Aichi-ken
  - Nagoya University Hospital /ID# 152709, Nagoya, Aichi-ken
  - Nagoya City University Hospital /ID# 151950, Nagoya, Aichi-ken
  - Toyohashi Municipal Hospital /ID# 171457, Toyohashi, Aichi-ken
  - Ieda Hospital /ID# 157781, Toyota-shi, Aichi-ken
  - Hirosaki National Hospital /ID# 152763, Hirosaki-shi, Aomori
  - Tokatsu Tsujinaka Hospital /ID# 214962, Abiko-shi, Chiba
  - Tsujinaka Hospital Kashiwanoha /ID# 209130, Kashiwa-shi, Chiba
  - Toho University Sakura Medical Center /ID# 151936, Sakura-shi, Chiba
  - Juntendo University Urayasu Hospital /ID# 208781, Urayasu-shi, Chiba
  - Fukui Prefectural Hospital /ID# 210448, Fukui-shi, Fukui
  - Fukuoka University Chikushi Hospital /ID# 152628, Chikushino-shi, Fukuoka
  - Saiseikai Fukuoka Genaral Hospital /ID# 209479, Fukuoka, Fukuoka
  - Kyushu University Hospital /ID# 152526, Fukuoka, Fukuoka
  - Kitakyushu Municipal Med Ctr /ID# 152588, Kitakyushu, Fukuoka
  - Kurume University Hospital /ID# 151976, Kurume-shi, Fukuoka
  - Ogaki Municipal Hospital /ID# 208225, Ogaki-shi, Gifu
  - NHO Fukuyama Medical Center /ID# 206293, Fukuyama-shi, Hiroshima
  - Hiroshima University Hospital /ID# 151951, Hiroshima, Hiroshima
  - Asahikawa Medical University Hospital /ID# 170289, Asahikawa-shi, Hokkaido
  - Obihiro kosei Hospital /ID# 210412, Obihiro-shi, Hokkaido
  - Sapporo Tokushukai Hospital /ID# 209397, Sapporo, Hokkaido
  - Hokkaido P.W.F.A.C. Sapporo-Kosei General Hospital /ID# 151506, Sapporo, Hokkaido
  - Sapporo Medical University Hospital /ID# 206492, Sapporo, Hokkaido
  - Sapporo Higashi Tokushukai Hospital /ID# 208487, Sapporo, Hokkaido
  - Aoyama Clinic /ID# 152049, Kobe, Hyōgo
  - Hyogo College of Medicine College Hospital /Id# 152434, Nishinomiya-shi, Hyōgo
  - National Hospital Organization Mito Medical Center /ID# 152631, Higashi Ibaraki-gun, Ibaraki
  - Kanazawa University Hospital /ID# 205099, Kanazawa, Ishikawa-ken
  - Iwate Medical University Uchimaru Medical Center /ID# 203411, Morioka, Iwate
  - Imamura General Hospital /ID# 227134, Kagoshima, Kagoshima-ken
  - Idzuro Imamura Hospital /ID# 206024, Kagoshima, Kagoshima-ken
  - Sameshima Hospital /ID# 206672, Kagoshima, Kagoshima-ken
  - St. Marianna University School of Medicine Hospital /ID# 208654, Kawasaki-shi, Kanagawa
  - Showa University Fujigaoka Hospital /ID# 208222, Yokohama, Kanagawa
  - Yokohama City University Medical Center /ID# 169899, Yokohama, Kanagawa
  - Japanese Red Cross Kyoto Daiichi Hosital /ID# 152359, Kyoto, Kyoto
  - Kyoto University Hospital /ID# 211758, Kyoto, Kyoto
  - Mie University Hospital /ID# 205362, Tsu, Mie-ken
  - Yokkaichi Hazu Medical Center /ID# 214347, Yokkaichi-shi, Mie-ken
  - National Hospital Organization Sendai Medical Center /ID# 209527, Sendai, Miyagi
  - NHO Nagasaki Medical Center /ID# 209531, Omura-shi, Nagasaki
  - Kenseikai Dongo Hospital /ID# 208100, Yamatotakada-shi, Nara
  - Saiseikai Niigata Hospital /ID# 209916, Niigata, Niigata
  - Niigata University Medical & Dental Hospital /ID# 218048, Niigata, Niigata
  - Ishida Clinic of IBD and Gastroenterology /ID# 210117, Ōita, Oita Prefecture
  - Chikuba Hospital for Proctological and Gastrointestinal Diseases /ID# 157821, Kurashiki-shi, Okayama-ken
  - Okayama University Hospital /ID# 217923, Okayama, Okayama-ken
  - Kinshukai Infusion Clinic /ID# 207864, Osaka, Osaka
  - Kitano Hospital /ID# 210395, Osaka, Osaka
  - Osaka City General Hospital /ID# 152704, Osaka, Osaka
  - Japanese Red Cross Osaka Hospital /ID# 209476, Osaka, Osaka
  - Osaka City University Hospital /ID# 152682, Osaka, Osaka
  - Toyonaka Municipal Hospital /ID# 217079, Toyonaka-shi, Osaka
  - Saga University Hospital /ID# 209268, Saga, Saga-ken
  - Saitama Medical Center /ID# 152031, Kawagoe-shi, Saitama
  - Tokitokai Tokito clinic /ID# 152677, Saitama-shi, Saitama
  - National Hospital Organization Higashi-Ohmi General Medical Center /ID# 210709, Higashi-ohmi-shi, Shiga
  - Shimane University Hospital /ID# 208899, Izumo-shi, Shimane
  - Hamamatsu University Hospital /ID# 205708, Hamamatsu, Shizuoka
  - NHO Shizuoka Medical Center /ID# 163572, Sunto-gun, Shizuoka
  - Tokyo Medical And Dental University Hospital /ID# 152016, Bunkyo-ku, Tokyo
  - St.Luke's International Hospital /ID# 208074, Chuo-ku, Tokyo
  - Tokai University Hachioji Hospital /ID# 152587, Hachioji-shi, Tokyo
  - Teikyo University Hospital /ID# 208897, Itabashi-ku, Tokyo
  - Kitasato University Kitasato Institute Hospital /ID# 152686, Minato-ku, Tokyo
  - Kyorin University Hospital /ID# 153194, Mitaka-shi, Tokyo
  - Center Hospital of the National Center for Global Health and Medicine /ID# 209267, Shinjuku-ku, Tokyo
  - Tokyo Women's Medical University Hospital /ID# 205977, Shinjuku-ku, Tokyo
  - Yamagata University Hospital /ID# 171454, Yamagata, Yamagata
  - Tokuyama Central Hospital /ID# 216993, Shunan-shi, Yamaguchi
  - Yamanashi Prefectural Central Hospital /ID# 151908, Kofu, Yamanashi
  - Shoyukai Fujita Gastroenterological Hospital /ID# 216492, Takatsuki-shi
- Latvia (2):
  - Pauls Stradins Clinical University Hospital /ID# 151409, Riga
  - Riga East Clinical University Hospital /ID# 150354, Riga
- Lithuania (4):
  - Hospital of Lithuanian University of Health Sciences Kaunas Clinics /ID# 150357, Kaunas
  - Klaipeda Seamens Hospital /ID# 154319, Klaipėda
  - Klaipeda University Hospital /ID# 158862, Klaipėda
  - Vilnius University Hospital /ID# 154318, Vilnius
- Malaysia (4):
  - Hospital Sultanah Bahiyah /ID# 151687, Alor Star, Kedah
  - Universiti Kebangsaan Malaysia (UKM) Medical Centre /ID# 151689, Kuala Lumpur, Selangor
  - Hospital Ampang /ID# 151298, Ampang
  - Uni Malaya MC /ID# 150359, Kuala Lumpur
- Mexico (3):
  - Morales Vargas Centro de Investigacion S.C. /ID# 211325, León, Guanajuato
  - Clinica de Investigacion en Reumatologia y Obesidad S.C. /ID# 150710, Guadalajara, Jalisco
  - Centro Regiomontano de Estudios Clínicos ROMA S.C /ID# 150256, Monterrey, Nuevo León
- Netherlands (5):
  - Radboud Universitair Medisch Centrum /ID# 151700, Nijmegen, Gelderland
  - Erasmus Medisch Centrum /ID# 150308, Rotterdam, South Holland
  - Academisch Medisch Centrum /ID# 150647, Amsterdam
  - Leids Universitair Medisch Centrum /ID# 152624, Leiden
  - Universitair Medisch Centrum Utrecht /ID# 152775, Utrecht
- Norway (2):
  - Akershus universitetssykehus /ID# 150317, Nordbyhagen, Akershus
  - Universitetssykehuset Nord-Norge /ID# 152835, Tromsø, Troms
- Poland (7):
  - Gastromed /Id# 216197, Torun, Kuyavian-Pomeranian Voivodeship
  - Centrum Zdrowia MDM /ID# 150351, Warsaw, Masovian Voivodeship
  - Centralny Szpital Kliniczny MSWiA w Warszawie /ID# 150580, Warsaw, Masovian Voivodeship
  - Centrum Medyczne Reuma Park /ID# 150349, Warsaw, Masovian Voivodeship
  - NZOZ Vivamed /ID# 216742, Warsaw, Masovian Voivodeship
  - Instytut Pomnik - Centrum Zdrowia Dziecka /ID# 215732, Warsaw, Masovian Voivodeship
  - Endoskopia Sp. z o.o. /ID# 150765, Sopot, Pomeranian Voivodeship
- Portugal (8):
  - Hospital da Senhora da Oliveira Guimaraes, EPE /ID# 151607, Guimarães, Braga District
  - Centro Hospitalar de Entre Douro e Vouga /ID# 152335, Santa Maria DA Feira, Porto District
  - Unidade Local de Saúde do Alto Minho, EPE - Hospital Conde de Bertiandos /ID# 151609, Ponte de Lima, Viana do Castelo District
  - Hospital Garcia de Orta, EPE /ID# 151613, Almada
  - CCA Braga - Hospital de Braga /ID# 151608, Braga
  - Centro Hospitalar Universitario Lisboa Central, EPE - Hospital dos Capuchos /ID# 151611, Lisbon
  - Centro Hospitalar Universitário de Lisboa Norte, EPE - Hospital de Santa Maria /ID# 151606, Lisbon
  - Centro Hospitalar Universitario de Sao Joao, EPE /ID# 151610, Porto
- School of Medicine University of Puerto Rico-Medical Science Campus /ID# 150358, San Juan, Puerto Rico
- Russia (11):
  - Immanuel Kant Baltic Federal University /ID# 200719, Kaliningrad, Kaliningrad Oblast
  - NW State Medical Univ na Mechn /ID# 169322, Saint Petersburg, Leningradskaya Oblast'
  - Perm Clinical Center of the Federal Medical and Biological Agency /ID# 150386, Perm, Permskiy Kray
  - Medical Company Hepatolog /ID# 200197, Samara, Samara Oblast
  - LLC Novaya Klinika /ID# 208107, Pyatigorsk, Stavropol Kray
  - Kazan State Medical University /ID# 166042, Kazan', Tatarstan, Respublika
  - Olla-Med Clinic /ID# 215332, Moscow
  - City Clinical Hospital #24 /ID# 150395, Moscow
  - Republican hospital named after V.A. Baranov /ID# 206506, Petrozavodsk
  - Euromedservice /ID# 203800, Pushkin
  - Duplicate_Stavropol State Medical Univ /ID# 150387, Stavropol
- Serbia (8):
  - Clinical Hosp Center Zvezdara /ID# 150427, Belgrade, Beograd
  - Military Medical Academy /ID# 150429, Belgrade, Beograd
  - University Clinical Center Serbia /ID# 150428, Belgrade, Beograd
  - Clin Hosp Ctr Bezanijska Kosa /ID# 150426, Belgrade, Beograd
  - University Clinical Center of Nis /ID# 151903, Niš, Nisavski Okrug
  - University Clinical Center Kragujevac /ID# 150430, Kragujevac, Sumadijski Okrug
  - Clinical Center Vojvodina /ID# 150764, Novi Sad, Vojvodina
  - General Hospital Leskovac /ID# 217880, Leskovac
- Singapore (3):
  - National University Hospital /ID# 150453, Singapore
  - Gleneagles Medical Centre /ID# 206018, Singapore
  - Tan Tock Seng Hospital /ID# 150443, Singapore
- Slovakia (6):
  - Fakultna nemocnica s poliklinikou F.D. Roosevelta Banska Bystrica /ID# 150868, Banská Bystrica
  - Medak s.r.o. /ID# 150480, Bratislava
  - Slovak Research Center Team Me /ID# 150257, Ilava
  - B+B MED, s.r.o. /ID# 150471, Košice
  - Fakultna nemocnica s poliklinikou Nove Zamky /ID# 211370, Nové Zámky
  - GASTRO I., s.r.o. /ID# 150472, Prešov
- South Africa (8):
  - MD Search /ID# 167293, Boksburg North, Gauteng
  - Clinresco Centers /ID# 163622, Johannesburg, Gauteng
  - Lenasia Clinical Trial Centre /ID# 214344, Johannesburg, Gauteng
  - Wits Clinical Research , Wits Health Consortium (PTY) Ltd /ID# 150785, Johannesburg, Gauteng
  - Wits Clinical Research Site /ID# 150496, Johannesburg, Gauteng
  - Kingsbury Hospital /ID# 150497, Cape Town, Western Cape
  - Private Practice Dr MN Rajabally /ID# 155144, Cape Town, Western Cape
  - Spoke Research Inc /ID# 162202, CAPE TOWN Milnerton, Western Cape
- South Korea (10):
  - Hayang University GuriHospital /ID# 150344, Guri-si, Gyeonggido
  - CHA University Bundang Medical Center /ID# 159479, Seongnam-si, Gyeonggido
  - The Catholic University of Korea, ST. Vincent's Hospital /ID# 150347, Suwon, Gyeonggido
  - Kangbuk Samsung Hospital /ID# 150348, Seoul, Seoul Teugbyeolsi
  - Yonsei University Health System Severance Hospital /ID# 159478, Seoul, Seoul Teugbyeolsi
  - Dong-A University Hospital /ID# 159480, Busan
  - Pusan National University Hospital /ID# 159481, Busan
  - Yeungnam University Medical Center /ID# 150345, Daegu
  - Asan Medical Center /ID# 150900, Seoul
  - Samsung Medical Center /ID# 150346, Seoul
- Spain (10):
  - Hospital Clínico Universitario de Santiago-CHUS /ID# 151065, Santiago de Compostela, A Coruna
  - Hospital Unversitario Marques de Valdecilla /ID# 216620, Santander, Cantabria
  - Hospital Universitario Dr. Negrin /ID# 203937, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Universitario A Coruna - CHUAC /ID# 203911, A Coruña
  - Hospital Clinic de Barcelona /ID# 150612, Barcelona
  - Hospital Universitario Reina Sofia /ID# 151066, Córdoba
  - Hospital Universitario Ramon y Cajal /ID# 151067, Madrid
  - Hospital Universitario La Paz /ID# 214539, Madrid
  - Hospital Universitario de Salamanca /ID# 150509, Salamanca
  - Hospital Universitario y Politecnico La Fe /ID# 150611, Valencia
- Sahlgrenska University Hospital /ID# 151496, Gothenburg, Västra Götaland County, Sweden
- Switzerland (4):
  - Universitätsspital Basel /ID# 161731, Basel, Canton of Basel-City
  - Kantonsspital St. Gallen /ID# 152599, Sankt Gallen, Canton of St. Gallen
  - Universitätsspital Zürich /ID# 152591, Zurich, Canton of Zurich
  - Inselspital, Universitätsspital Bern /ID# 152590, Bern
- Taiwan (6):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital /ID# 150575, Kaohsiung City
  - Chung Shan Medical University Hospital /ID# 150573, Taichung
  - China Medical University Hospital /ID# 150571, Taichung
  - National Cheng Kung University Hospital /ID# 151749, Tainan
  - National Taiwan University Hospital /ID# 150574, Taipei
  - Taipei Veterans General Hosp /ID# 151748, Taipei
- Turkey (Türkiye) (6):
  - Erciyes University Medical Fac /ID# 150129, Melikgazi, Kayseri
  - Istanbul University-Cerrahpasa, Cerrahpasa Medical Faculty /ID# 150125, Istanbul
  - Umraniye Training and Res Hosp /ID# 162659, Istanbul
  - Marmara University Medical Fac /ID# 213969, Istanbul
  - Mersin University Medical /ID# 157849, Mersin
  - Gazi Universitesi Tip Fakultes /ID# 150127, Yenimahalle
- Ukraine (10):
  - Medical Center of the "Health /ID# 151274, Vinnytsia, Vinnytsia Oblast
  - Municipal Enterprise "I.I. Mechnikov Dnipropetrovsk Regional Clinical Hospital" /ID# 207723, Dnipro
  - CNCE of Kharkiv Regional Council Regional Clinical Hospital /ID# 206940, Kharkiv
  - PE PMC Acinus, Medical and Diagnostic Center /ID# 217216, Kropyvnytskyi
  - Kyiv Municipal Clinical Hospital #18 /ID# 150372, Kyiv
  - Medical Center CONSILIUM MEDICAL /ID# 217446, Kyiv
  - CNPE of Kyiv Regional Council Kyiv Regional Hospital /ID# 217372, Kyiv
  - Lviv Regional Clinical Hospital /ID# 150375, Lviv
  - Municipal Non-Commercial Enterprise Odesa Regional Clinical Hospital of the Od /ID# 151275, Odesa
  - CNE Vinnytsya Regional Clinical Hospital named after N.I.Pirogov /ID# 216297, Vinnytsia
- United Kingdom (8):
  - Royal Devon and Exeter NHS Trust Hospital /ID# 150379, Exeter, Devon
  - Hampshire Hospitals NHS Foundation Trust /ID# 150380, Basingstoke, Essex
  - Barts Health NHS Trust /ID# 150384, London, London, City of
  - NHS Greater Glasgow and Clyde /ID# 163787, Glasgow, Scotland
  - Royal United Hospitals Bath /ID# 151532, Bath
  - University Hospitals Birmingham NHS Foundation Trust /ID# 150382, Birmingham
  - Calderdale and Huddersfield NHS Foundation Trust /ID# 217658, Huddersfield
  - St George's University Hospitals NHS Foundation Trust /ID# 208374, Tooting

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing, please refer to the link below.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Use Agreement (DUA). For more information on the process, or to submit a request, visit the following link.
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Burmester GR, Deodhar A, Irvine AD, Panaccione R, Winthrop KL, Vleugels RA, Levy G, Suravaram S, Palac H, Wegrzyn L, Ford S, Meerwein S, Guttman-Yassky E. Safety Profile of Upadacitinib: Descriptive Analysis in Over 27,000 Patient-Years Across Rheumatoid Arthritis, Psoriatic Arthritis, Axial Spondyloarthritis, Atopic Dermatitis, and Inflammatory Bowel Disease. Adv Ther. 2025 Oct;42(10):5215-5237. doi: 10.1007/s12325-025-03328-y. Epub 2025 Aug 28. PMID 40875187
- [Derived] Panes J, Dubinsky MC, Ishiguro Y, Shukla N, Dubcenco E, Remple V, Sharma D, Panaccione R. Achievement of long-term treatment goals in upadacitinib-treated patients with moderately to severely active ulcerative colitis: a post hoc analysis of phase 3 trial data. J Crohns Colitis. 2025 Jul 3;19(7):jjaf095. doi: 10.1093/ecco-jcc/jjaf095. PMID 40488552
- [Derived] Panaccione R, Danese S, Zhou W, Klaff J, Ilo D, Yao X, Levy G, Higgins PDR, Loftus EV Jr, Chen S, Gonzalez YS, Leonard C, Hebuterne X, Lindsay JO, Cao Q, Nakase H, Colombel JF, Vermeire S. Efficacy and safety of upadacitinib for 16-week extended induction and 52-week maintenance therapy in patients with moderately to severely active ulcerative colitis. Aliment Pharmacol Ther. 2024 Feb;59(3):393-408. doi: 10.1111/apt.17816. Epub 2023 Nov 27. PMID 38010661
- [Derived] Raine T, Ishiguro Y, Rubin DT, Finney-Hayward T, Vladea R, Liu J, Phillips C, Cheng E, Targownik L, Loftus EV Jr. Impact of Baseline Corticosteroid Use on the Efficacy and Safety of Upadacitinib in Patients with Ulcerative Colitis: A Post Hoc Analysis of the Phase 3 Clinical Trial Programme. J Crohns Colitis. 2024 May 31;18(5):695-707. doi: 10.1093/ecco-jcc/jjad190. PMID 37942921
- [Derived] Vermeire S, Danese S, Zhou W, Ilo D, Klaff J, Levy G, Yao X, Chen S, Sanchez Gonzalez Y, Hebuterne X, Lindsay JO, Higgins PDR, Cao Q, Nakase H, Colombel JF, Loftus EV Jr, Panaccione R. Efficacy and safety of upadacitinib maintenance therapy for moderately to severely active ulcerative colitis in patients responding to 8 week induction therapy (U-ACHIEVE Maintenance): overall results from the randomised, placebo-controlled, double-blind, phase 3 maintenance study. Lancet Gastroenterol Hepatol. 2023 Nov;8(11):976-989. doi: 10.1016/S2468-1253(23)00208-X. Epub 2023 Sep 9. PMID 37683686
- [Derived] Parkes G, Ungaro RC, Danese S, Abreu MT, Arenson E, Zhou W, Ilo D, Laroux FS, Deng H, Sanchez Gonzalez Y, Peyrin-Biroulet L. Correlation of mucosal healing endpoints with long-term clinical and patient-reported outcomes in ulcerative colitis. J Gastroenterol. 2023 Oct;58(10):990-1002. doi: 10.1007/s00535-023-02013-7. Epub 2023 Jul 25. PMID 37490069
- [Derived] Loftus EV Jr, Ananthakrishnan AN, Lee WJ, Gonzalez YS, Fitzgerald KA, Wallace K, Zhou W, Litcher-Kelly L, Ollis SB, Su S, Danese S. Content Validity and Psychometric Evaluation of the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) in Patients with Crohn's Disease and Ulcerative Colitis. Pharmacoecon Open. 2023 Sep;7(5):823-840. doi: 10.1007/s41669-023-00419-w. Epub 2023 Jun 9. PMID 37296268
- [Derived] Danese S, Tran J, D'Haens G, Rubin DT, Aoyama N, Zhou W, Ilo D, Yao X, Sanchez Gonzalez Y, Panaccione R. Upadacitinib Induction and Maintenance Therapy Improves Abdominal Pain, Bowel Urgency, and Fatigue in Patients With Ulcerative Colitis: A Post Hoc Analysis of Phase 3 Data. Inflamm Bowel Dis. 2023 Nov 2;29(11):1723-1729. doi: 10.1093/ibd/izad016. PMID 36790041
- [Derived] Panes J, Loftus EV, Higgins PDR, Lindsay JO, Zhou W, Yao X, Ilo D, Phillips C, Tran J, Sanchez Gonzalez Y, Vermeire S. Induction and Maintenance Treatment With Upadacitinib Improves Health-Related Quality of Life in Patients With Moderately to Severely Active Ulcerative Colitis: Phase 3 Study Results. Inflamm Bowel Dis. 2023 Sep 1;29(9):1421-1430. doi: 10.1093/ibd/izac260. PMID 36645051
- [Derived] Ponce-Bobadilla AV, Stodtmann S, Eckert D, Zhou W, Liu W, Mohamed MF. Upadacitinib Population Pharmacokinetics and Exposure-Response Relationships in Ulcerative Colitis Patients. Clin Pharmacokinet. 2023 Jan;62(1):101-112. doi: 10.1007/s40262-022-01191-6. Epub 2022 Dec 26. PMID 36571701
- [Derived] Loftus EV Jr, Colombel JF, Takeuchi K, Gao X, Panaccione R, Danese S, Dubinsky M, Schreiber S, Ilo D, Finney-Hayward T, Zhou W, Phillips C, Gonzalez YS, Shu L, Yao X, Zhou Q, Vermeire S. Upadacitinib Therapy Reduces Ulcerative Colitis Symptoms as Early as Day 1 of Induction Treatment. Clin Gastroenterol Hepatol. 2023 Aug;21(9):2347-2358.e6. doi: 10.1016/j.cgh.2022.11.029. Epub 2022 Dec 1. PMID 36464141
- [Derived] Danese S, Vermeire S, Zhou W, Pangan AL, Siffledeen J, Greenbloom S, Hebuterne X, D'Haens G, Nakase H, Panes J, Higgins PDR, Juillerat P, Lindsay JO, Loftus EV Jr, Sandborn WJ, Reinisch W, Chen MH, Sanchez Gonzalez Y, Huang B, Xie W, Liu J, Weinreich MA, Panaccione R. Upadacitinib as induction and maintenance therapy for moderately to severely active ulcerative colitis: results from three phase 3, multicentre, double-blind, randomised trials. Lancet. 2022 Jun 4;399(10341):2113-2128. doi: 10.1016/S0140-6736(22)00581-5. Epub 2022 May 26. PMID 35644166
- [Derived] Sandborn WJ, Ghosh S, Panes J, Schreiber S, D'Haens G, Tanida S, Siffledeen J, Enejosa J, Zhou W, Othman AA, Huang B, Higgins PDR. Efficacy of Upadacitinib in a Randomized Trial of Patients With Active Ulcerative Colitis. Gastroenterology. 2020 Jun;158(8):2139-2149.e14. doi: 10.1053/j.gastro.2020.02.030. Epub 2020 Feb 22. PMID 32092309
- See also: This clinical study may be evaluating a usage that is not currently FDA approved. Please see US Prescribing Information for approved uses. — https://www.rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Intent-to-treat (ITT) analysis set: Substudy 1 (all randomized participants who received at least one dose of study drug in Substudy 1); Substudy 2 (all randomized participants who received at least one dose of doubleblinded study drug in Part 1 and all participants who received at least one dose of upadacitinib 45 mg in Part 2); Substudy 3 (all participants who received at least one dose of study drug in Substudy 3)
Groups:
- SS3: M14-675 Clinical Responders: Participants in Study M14-675 (NCT03653026) who achieved clinical response defined by Adapted Mayo Score at Week 8 or Week 16 in that study and did not meet any study discontinuation criteria were eligible to enroll into Substudy 3. Participants were treated with a blinded treatment assignment (15 mg upadacitinib film-coated tablets once daily by mouth [QD], or 30 mg upadacitinib film-coated tablets QD, or placebo for upadacitinib film-coated tablets QD) for up to 52 weeks.
- SS3: Placebo: Participants who achieved clinical response in Substudy 1, Substudy 2, or Study M14-675 at either Week 8 or Week 16, while receiving upadacitinib 15, 30, or 45 mg QD and those who achieved clinical response while receiving upadacitinib 15 mg QD in Substudy 1 and were randomized to placebo QD in Substudy 3 for up to 52 weeks. In addition, participants who received double-blind placebo QD treatment for 8 weeks during Substudy 1, Substudy 2 Part 1, or Study M14-675 Part 1 and achieved clinical response at Week 8 continued to receive blinded placebo QD in Substudy 3 for up to 52 weeks.
- SS3: UPA 7.5 mg: Participants who received double-blinded treatment of upadacitinib 7.5 mg QD for 8 weeks during Substudy 1 and achieved clinical response at Week 8 continued to receive blinded treatment of upadacitinib 7.5 mg QD in Substudy 3 for up to 52 weeks.
- SS3: UPA 15 mg: Participants who achieved clinical response in Substudy 1, Substudy 2, or Study M14-675 at either Week 8 or Week 16, while receiving upadacitinib 15, 30, or 45 mg QD and those who achieved clinical response while receiving upadacitinib 15 mg QD in Substudy 1 and were randomized to upadacitinib 15 mg QD in Substudy 3 for up to 52 weeks. In addition, participants who received upadacitinib 45 mg QD in Induction Phase and did not achieve clinical response and received upadacitinib 45 mg QD in Extended Treatment in Substudy 2 Part 2 or in Study M14-675 Part 2 and achieved clinical response at Week 16 and were randomized to upadacitinib 15 mg QD in Substudy 3.
- SS3: UPA 30 mg: Participants who achieved clinical response in Substudy 1, Substudy 2, or Study M14-675 at either Week 8 or Week 16, while receiving upadacitinib 15, 30, or 45 mg QD and those who achieved clinical response while receiving upadacitinib 15 mg QD in Substudy 1 and were randomized to upadacitinib 30 mg QD in Substudy 3 for up to 52 weeks. In addition, participants who received upadacitinib 45 mg QD in Induction Phase and did not achieve clinical response and received upadacitinib 45 mg QD in Extended Treatment in Substudy 2 Part 2 or in Study M14-675 Part 2 and achieved clinical response at Week 16 and were randomized to upadacitinib 30 mg QD in Substudy 3.
Period: Substudy 1 and Substudy 2, Part 1
Arm/Group | SS1: Placebo | SS1: Upadacitinib 7.5 mg | SS1: Upadacitinib 15 mg | SS1: Upadacitinib 30 mg | SS1: Upadacitinib 45 mg | SS2: Placebo/Upadacitinib 45 mg | SS2: Upadacitinib 45 mg/Upadacitinib 45 mg | SS3: M14-675 Clinical Responders | SS3: Placebo | SS3: UPA 7.5 mg | SS3: UPA 15 mg | SS3: UPA 30 mg
Started | 46 | 47 | 49 | 117 | 123 | 155 | 319 | 446 | 0 | 0 | 0 | 0
Completed | 41 | 45 | 45 | 105 | 113 | 135 | 306 | 446 | 0 | 0 | 0 | 0
Not Completed | 5 | 2 | 4 | 12 | 10 | 20 | 13 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 3 | 1 | 3 | 5 | 4 | 9 | 6 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrew consent | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — COVID-19 Logistical Restrictions | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Other, not specified | 2 | 1 | 1 | 7 | 5 | 7 | 3 | 0 | 0 | 0 | 0 | 0
Period: Substudy 2, Part 2
Arm/Group | SS1: Placebo | SS1: Upadacitinib 7.5 mg | SS1: Upadacitinib 15 mg | SS1: Upadacitinib 30 mg | SS1: Upadacitinib 45 mg | SS2: Placebo/Upadacitinib 45 mg | SS2: Upadacitinib 45 mg/Upadacitinib 45 mg | SS3: M14-675 Clinical Responders | SS3: Placebo | SS3: UPA 7.5 mg | SS3: UPA 15 mg | SS3: UPA 30 mg
Started | 0 | 0 | 0 | 0 | 0 | 85 | 59 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 74 | 47 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 11 | 12 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrew consent | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — COVID-19 Logistical Restrictions | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Other, not specified | 0 | 0 | 0 | 0 | 0 | 4 | 8 | 0 | 0 | 0 | 0 | 0
Period: Substudy 3
Arm/Group | SS1: Placebo | SS1: Upadacitinib 7.5 mg | SS1: Upadacitinib 15 mg | SS1: Upadacitinib 30 mg | SS1: Upadacitinib 45 mg | SS2: Placebo/Upadacitinib 45 mg | SS2: Upadacitinib 45 mg/Upadacitinib 45 mg | SS3: M14-675 Clinical Responders | SS3: Placebo | SS3: UPA 7.5 mg | SS3: UPA 15 mg | SS3: UPA 30 mg
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 386 | 20 | 324 | 316
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 140 | 11 | 218 | 248
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 246 | 9 | 106 | 68
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 32 | 3 | 12 | 18
Not completed — Withdrew consent | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 1 | 4 | 9
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Not completed — COVID-19 Logistical Restrictions | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Other, not specified | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 202 | 5 | 89 | 39

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) analysis set: Substudy 1 (all randomized participants who received at least one dose of study drug in Substudy 1); Substudy 2 (all randomized participants who received at least one dose of doubleblinded study drug in Part 1 and all participants who received at least one dose of upadacitinib 45 mg in Part 2); Substudy 3 (all M14-675 participants who received at least one dose of study drug in Substudy 3)
Groups:
- Total: Total of all reporting groups
Arm/Group | SS1: Placebo | SS1: Upadacitinib 7.5 mg | SS1: Upadacitinib 15 mg | SS1: Upadacitinib 30 mg | SS1: Upadacitinib 45 mg | SS2: Placebo/Upadacitinib 45 mg | SS2: Upadacitinib 45 mg/Upadacitinib 45 mg | SS3: M14-675 Clinical Responders | Total
Number analyzed (Participants) | 46 | 47 | 49 | 117 | 123 | 155 | 319 | 446 | 1302
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.3 (13.29) | 41.7 (14.58) | 46.0 (13.58) | 42.9 (14.44) | 41.6 (14.19) | 44.3 (14.64) | 43.6 (14.04) | 42.1 (14.42) | 42.9 (14.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 24 | 19 | 47 | 44 | 58 | 121 | 170 | 500
  Male | 29 | 23 | 30 | 70 | 79 | 97 | 198 | 276 | 802
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 37 | 36 | 38 | 88 | 90 | 101 | 206 | 302 | 898
  Black or African American | 0 | 3 | 1 | 3 | 2 | 4 | 12 | 15 | 40
  Asian | 8 | 7 | 10 | 23 | 28 | 46 | 95 | 124 | 341
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
  Multiple | 1 | 1 | 0 | 2 | 3 | 2 | 5 | 3 | 17
Average Stool Frequency Subscore [Mean (Standard Deviation); unit: units on a scale] — Participants recorded stool frequency using an electronic subject diary on a daily basis. The stool frequency subscore (SFS) ranges from 0 to 3 according to the following scale:
  Score 0: Normal number of stools
  Score 1: 1 to 2 stools more than normal
  Score 2: 3 to 4 stools more than normal
  Score 3: 5 or more stools more than normal Population: Participants with available data
  units on a scale
    number analyzed (Participants) | 46 | 47 | 49 | 117 | 122 | 155 | 318 | 445 | 1299
    (all) | 2.56 (0.667) | 2.62 (0.600) | 2.68 (0.565) | 2.61 (0.613) | 2.58 (0.648) | 2.52 (0.668) | 2.60 (0.624) | 2.55 (0.623) | 2.58 (0.628)
Average Rectal Bleeding Subscore [Mean (Standard Deviation); unit: units on a scale] — Participants recorded rectal bleeding in an electronic subject diary on a daily basis. The rectal bleeding subscore ranges from 0 to 3 according to the following scale:
  Score 0: No blood seen
  Score 1: Streaks of blood with stool less than half the time
  Score 2: Obvious blood with stool most of the time
  Score 3: Blood alone passed Population: Participants with available data
  units on a scale
    number analyzed (Participants) | 46 | 47 | 49 | 117 | 122 | 155 | 318 | 445 | 1299
    (all) | 1.66 (1.034) | 1.61 (1.027) | 1.55 (0.915) | 1.51 (0.975) | 1.49 (0.960) | 1.76 (0.994) | 1.71 (1.046) | 1.77 (0.990) | 1.68 (1.003)
Average Endoscopy Subscore [Mean (Standard Deviation); unit: units on a scale] — Findings on endoscopy were scored according to the following:
  Score 0: Normal or inactive disease
  Score 1: Mild disease (erythema, decreased vascular pattern)
  Score 2: Moderate disease (marked erythema, lack of vascular pattern, any friability, erosions)
  Score 3: Severe disease (spontaneous bleeding, ulceration)
  units on a scale | 2.8 (0.43) | 2.8 (0.40) | 2.8 (0.39) | 2.7 (0.47) | 2.7 (0.48) | 2.7 (0.47) | 2.7 (0.46) | 2.7 (0.47) | 2.7 (0.46)
Previous Biologic Use [Count of Participants; unit: Participants] — Population: Participants with available data
  Participants
    Yes: number analyzed (Participants) | 46 | 47 | 49 | 117 | 123 | 0 | 0 | 0 | 382
    Yes | 35 | 36 | 38 | 87 | 92 |  |  |  | 288
    No: number analyzed (Participants) | 46 | 47 | 49 | 117 | 123 | 0 | 0 | 0 | 382
    No | 11 | 11 | 11 | 30 | 31 |  |  |  | 94
Biologic-inadequate Responder (Bio-IR) Status [Count of Participants; unit: Participants] — Biologic-inadequate responders (Bio-IR) are defined as participants who had inadequate response, loss of response, or intolerance to biologic therapy.
  Non-biologic-inadequate responders (non-bio-IR) are defined as participants who had inadequate response, loss of response, or intolerance to conventional therapy but had not failed biologic therapy. Population: Participants with available data
  Participants
    Bio-IR: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 155 | 319 | 446 | 920
    Bio-IR |  |  |  |  |  | 79 | 168 | 221 | 468
    Non-Bio-IR: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 155 | 319 | 446 | 920
    Non-Bio-IR |  |  |  |  |  | 76 | 151 | 225 | 452
Baseline Corticosteroid Use [Count of Participants; unit: Participants]
  Yes | 26 | 24 | 27 | 51 | 53 | 62 | 124 | 173 | 540
  No | 20 | 23 | 22 | 66 | 70 | 93 | 195 | 273 | 762

OUTCOME MEASURES:

1. Primary Outcome: Substudy 1: Percentage Of Participants Who Achieved Clinical Remission Per Adapted Mayo Score at Week 8
Description: The Adapted Mayo Score is a composite score of UC disease activity based on the following 3 subscores:
  1. Stool frequency subscore (SFS), scored from 0 (normal number of stools) to 3 (5 or more stools more than normal)
  2. Rectal bleeding subscore (RBS), scored from 0 (no blood seen) to 3 (blood alone passed)
  3. Endoscopic subscore, scored from 0 (normal or inactive disease) to 3 (severe disease, spontaneous bleeding, ulceration)
  The overall Adapted Mayo score ranges from 0 to 9 where higher scores represent more severe disease.
  For Substudy 1, clinical remission is defined as SFS ≤ 1, RBS of 0, and endoscopic subscore ≤ 1.
Time Frame: At Week 8
Population: SS1 main population (ITT1A): those randomized to ≥1 dose of study drug during the initial part of SS1. Non-responder imputation (NRI) was used to impute missing values.
Measure: Number; unit: percentage of participants
Arm/Group | SS1: Placebo | SS1: Upadacitinib 7.5 mg | SS1: Upadacitinib 15 mg | SS1: Upadacitinib 30 mg | SS1: Upadacitinib 45 mg
Number analyzed (Participants) | 46 | 47 | 49 | 52 | 56
percentage of participants | 0 | 8.5 | 14.3 | 13.5 | 21.4
Statistical Analysis 1: Comparison: SS1: Placebo vs SS1: Upadacitinib 7.5 mg; Substudy 1: Upadacitinib 7.5 mg vs Placebo; Test type: Superiority; p = 0.049, Cochran-Mantel-Haenszel — The primary and ranked secondary efficacy endpoints were tested with multiplicity adjustment using a fixed-sequence multiple testing procedure to ensure a strong control of family-wise type I error rate at significance level alpha = 0.05 (2-sided); Stratified by previous biologic use, baseline corticosteroid use and baseline Adapted Mayo score (≤ 7 and > 7); Adjusted risk difference (%) = 8.4, 95% CI 2-sided [0.0 to 16.8] — Difference = Upadacitinib 7.5 mg - Placebo
Statistical Analysis 2: Comparison: SS1: Placebo vs SS1: Upadacitinib 15 mg; Substudy 1: Upadacitinib 15 mg vs Placebo; Test type: Superiority; p = 0.010, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Stratified by previous biologic use, baseline corticosteroid use and baseline Adapted Mayo score (≤ 7 and > 7); Adjusted risk difference (%) = 13.5, 95% CI 2-sided [3.3 to 23.8] — Difference = Upadacitinib 15 mg - Placebo
Statistical Analysis 3: Comparison: SS1: Placebo vs SS1: Upadacitinib 30 mg; Substudy 1: Upadacitinib 30 mg vs Placebo; Test type: Superiority; p = 0.007, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Stratified by previous biologic use, baseline corticosteroid use and baseline Adapted Mayo score (≤ 7 and > 7); Adjusted risk difference (%) = 13.8, 95% CI 2-sided [3.8 to 23.9] — Difference = Upadacitinib 30 mg - Placebo
Statistical Analysis 4: Comparison: SS1: Placebo vs SS1: Upadacitinib 45 mg; Substudy 1: Upadacitinib 45 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Stratified by previous biologic use, baseline corticosteroid use and baseline Adapted Mayo score (≤ 7 and > 7); Adjusted risk difference (%) = 21.1, 95% CI 2-sided [8.6 to 33.6] — Difference = Upadacitinib 45 mg - Placebo

2. Primary Outcome: Substudy 2: Percentage Of Participants Who Achieved Clinical Remission Per Adapted Mayo Score at Week 8
Description: The Adapted Mayo Score is a composite score of UC disease activity based on the following 3 subscores:
  1. Stool frequency subscore (SFS), scored from 0 (normal number of stools) to 3 (5 or more stools more than normal)
  2. Rectal bleeding subscore (RBS), scored from 0 (no blood seen) to 3 (blood alone passed)
  3. Endoscopic subscore, scored from 0 (normal or inactive disease) to 3 (severe disease, spontaneous bleeding, ulceration)
  The overall Adapted Mayo score ranges from 0 to 9 where higher scores represent more severe disease.
  For Substudy 2, clinical remission is defined as SFS ≤ 1 and not greater than Baseline, RBS of 0, and endoscopic subscore ≤ 1. In Substudy 2, evidence of friability during endoscopy in participants with otherwise "mild" endoscopic activity conferred an endoscopic subscore of 2.
Time Frame: At Week 8
Population: SS2, Part 1 population (ITT1): all randomized participants in the 8-week double-blind induction period who received ≥1 dose of study drug. NRI incorporating multiple imputation (MI) to handle missing data due to COVID-19 (NRI-C) was used for SS2, with participants analyzed according to treatment groups to which they were randomized.
Measure: Number; unit: percentage of participants
Groups:
- SS2: Placebo: During the Substudy 2 Part 1 induction period, participants received placebo for upadacitinib film-coated tablets once daily by mouth (QD) for 8 weeks.
- SS2: Upadacitinib 45 mg: During the Substudy 2 Part 1 induction period, participants received 45 mg upadacitinib film-coated tablets once daily by mouth (QD) for 8 weeks.
Arm/Group | SS2: Placebo | SS2: Upadacitinib 45 mg
Number analyzed (Participants) | 154 | 319
percentage of participants | 4.8 | 26.1
Statistical Analysis 1: Comparison: SS2: Placebo vs SS2: Upadacitinib 45 mg; Substudy 2: Upadacitinib 45 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Stratified by bio-IR status (bio-IR vs. non-bio-IR), Baseline corticosteroid use (yes vs. no) and Baseline Adapted Mayo score (≤ 7 vs. > 7); Adjusted risk difference (%) = 21.6, 95% CI 2-sided [15.8 to 27.4] — Difference = Upadacitinib 45 mg - Placebo

3. Primary Outcome: Substudy 3: Percentage Of Participants Who Achieved Clinical Remission Per Adapted Mayo Score at Week 52
Description: The Adapted Mayo Score is a composite score of UC disease activity based on the following 3 subscores:
  1. Stool frequency subscore (SFS), scored from 0 (normal number of stools) to 3 (5 or more stools more than normal).
  2. Rectal bleeding subscore (RBS), scored from 0 (no blood seen) to 3 (blood alone passed).
  3. Endoscopic subscore, scored from 0 (normal or inactive disease) to 3 (severe disease, spontaneous bleeding, ulceration).
  The overall Adapted Mayo score ranges from 0 to 9 where higher scores represent more severe disease.
  For Substudy 3, clinical remission is defined as SFS ≤ 1 and not greater than Baseline, RBS of 0, and endoscopic subscore ≤ 1. In addition, evidence of friability during endoscopy in participants with otherwise "mild" endoscopic activity conferred an endoscopic subscore of 2.
Time Frame: At Week 52
Population: Substudy 3 ITT_A population: the first 451 upadacitinib 45 mg 8-week induction responders who were enrolled under the protocol for 52-week maintenance treatment period in Cohort 1. Non-responder imputation incorporating multiple imputation (MI) to handle missing data due to COVID-19 (NRI-C) was used to handle missing data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- SS3: Placebo: Participants who achieved clinical response in Substudy 1, Substudy 2, or Study M14-675 at Week 8, while receiving upadacitinib 15, 30, or 45 mg QD and were randomized to placebo QD in Substudy 3 for up to 52 weeks. In addition, participants who received double-blind placebo QD treatment for 8 weeks during Substudy 1, Substudy 2 Part 1, or Study M14-675 Part 1 and achieved clinical response at Week 8 continued to receive blinded placebo QD in Substudy 3 for up to 52 weeks.
- SS3: UPA 15 mg: Participants who achieved clinical response in Substudy 1, Substudy 2, or Study M14-675 at Week 8 while receiving upadacitinib 15, 30, or 45 mg QD and were randomized to upadacitinib 15 mg QD in Substudy 3 for up to 52 weeks
- SS3: UPA 30 mg: Participants who achieved clinical response in Substudy 1, Substudy 2, or Study M14-675 at Week 8 while receiving upadacitinib 15, 30, or 45 mg QD and were randomized to upadacitinib 30 mg QD in Substudy 3 for up to 52 weeks
Arm/Group | SS3: Placebo | SS3: UPA 15 mg | SS3: UPA 30 mg
Number analyzed (Participants) | 149 | 148 | 154
percentage of participants | 12.1 [6.9 to 17.4] | 42.3 [34.3 to 50.3] | 51.7 [43.6 to 59.8]
Statistical Analysis 1: Comparison: SS3: Placebo vs SS3: UPA 15 mg; Substudy 3: Upadacitinib 15 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Stratified by Bio-IR (Bio-IR/Non-Bio-IR) at Baseline of Induction Study; clinical remission at Week 0 (yes/no); corticosteroid use at Week 0 (yes/no); Adjusted risk difference (%) = 30.7, 95% CI 2-sided [21.7 to 39.8] — Difference = Upadacitinib 15 mg - Placebo
Statistical Analysis 2: Comparison: SS3: Placebo vs SS3: UPA 30 mg; Substudy 3: Upadacitinib 30 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 3, analysis 1]; Adjusted risk difference (%) = 39.0, 95% CI 2-sided [29.7 to 48.2] — Difference = Upadacitinib 30 mg - Placebo

4. Secondary Outcome: Substudy 1: Percentage Of Participants With Endoscopic Improvement at Week 8
Description: Endoscopic improvement is defined as an endoscopic subscore of 0 or 1. Endoscopies were assessed by a blinded central reader and scored according to the following scale: 0 = Normal or inactive disease; 1 = Mild disease (erythema, decreased vascular pattern); 2 = Moderate disease (marked erythema, lack of vascular pattern, any friability, erosions); 3 = Severe disease (spontaneous bleeding, ulceration).
Time Frame: At Week 8
Population: The Substudy 1 main population (ITT1A) includes participants who were randomized to at least one dose (placebo or upadacitinib 7.5 mg, 15 mg, 30 mg, 45 mg) during the main (initial) part of Substudy 1. Non-responder imputation (NRI) was used to impute missing values for the ITT1A population.
Measure: Number; unit: percentage of participants
Arm/Group | SS1: Placebo | SS1: Upadacitinib 7.5 mg | SS1: Upadacitinib 15 mg | SS1: Upadacitinib 30 mg | SS1: Upadacitinib 45 mg
Number analyzed (Participants) | 46 | 47 | 49 | 52 | 56
percentage of participants | 2.2 | 14.9 | 30.6 | 26.9 | 35.7
Statistical Analysis 1: Comparison: SS1: Placebo vs SS1: Upadacitinib 7.5 mg; Substudy 1: Upadacitinib 7.5 mg vs Placebo; Test type: Superiority; p = 0.030, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Stratified by previous biologic use, baseline corticosteroid use and baseline Adapted Mayo score (≤ 7 and > 7); Adjusted risk difference (%) = 13.1, 95% CI 2-sided [1.2 to 25.0] — Difference = Upadacitinib 7.5 mg - Placebo
Statistical Analysis 2: Comparison: SS1: Placebo vs SS1: Upadacitinib 15 mg; Substudy 1: Upadacitinib 15 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Stratified by previous biologic use, baseline corticosteroid use and baseline Adapted Mayo score (≤ 7 and > 7); Adjusted risk difference (%) = 27.6, 95% CI 2-sided [13.1 to 42.1] — Difference = Upadacitinib 15 mg - Placebo
Statistical Analysis 3: Comparison: SS1: Placebo vs SS1: Upadacitinib 30 mg; Substudy 1: Upadacitinib 30 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Stratified by previous biologic use, baseline corticosteroid use and baseline Adapted Mayo score (≤ 7 and > 7); Adjusted risk difference (%) = 26.6, 95% CI 2-sided [12.3 to 40.8] — Difference = Upadacitinib 30 mg - Placebo
Statistical Analysis 4: Comparison: SS1: Placebo vs SS1: Upadacitinib 45 mg; Substudy 1: Upadacitinib 45 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Stratified by previous biologic use, baseline corticosteroid use and baseline Adapted Mayo score (≤ 7 and > 7); Adjusted risk difference (%) = 35.4, 95% CI 2-sided [19.2 to 51.7] — Difference = Upadacitinib 45 mg - Placebo

5. Secondary Outcome: Substudy 1: Percentage Of Participants Achieving Clinical Remission Per Full Mayo Score at Week 8
Description: The Mayo score is a tool designed to measure disease activity for ulcerative colitis. The Full Mayo score (FMS) ranges from 0 (normal or inactive disease) to 12 (severe disease) and is calculated as the sum of 4 subscores (stool frequency, rectal bleeding, endoscopy [confirmed by a central reader], and physician's global assessment), each of which ranges from 0 (normal) to 3 (severe disease). Negative changes indicate improvement. Clinical remission per FMS is defined as Mayo Score ≤ 2 and no individual subscore > 1.
Time Frame: At Week 8
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | SS1: Placebo | SS1: Upadacitinib 7.5 mg | SS1: Upadacitinib 15 mg | SS1: Upadacitinib 30 mg | SS1: Upadacitinib 45 mg
Number analyzed (Participants) | 46 | 47 | 49 | 52 | 56
percentage of participants | 0 | 10.6 | 10.2 | 11.5 | 19.6
Statistical Analysis 1: Comparison: SS1: Placebo vs SS1: Upadacitinib 7.5 mg; Substudy 1: Upadacitinib 7.5 mg vs Placebo; Test type: Superiority; p = 0.021, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Stratified by previous biologic use, baseline corticosteroid use and baseline Adapted Mayo score (≤ 7 and > 7); Adjusted risk difference (%) = 11.0, 95% CI 2-sided [1.7 to 20.4] — Difference = Upadacitinib 7.5 mg - Placebo
Statistical Analysis 2: Comparison: SS1: Placebo vs SS1: Upadacitinib 15 mg; Substudy 1: Upadacitinib 15 mg vs Placebo; Test type: Superiority; p = 0.024, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Stratified by previous biologic use, baseline corticosteroid use and baseline Adapted Mayo score (≤ 7 and > 7); Adjusted risk difference (%) = 9.6, 95% CI 2-sided [1.3 to 18.0] — Difference = Upadacitinib 15 mg - Placebo
Statistical Analysis 3: Comparison: SS1: Placebo vs SS1: Upadacitinib 30 mg; Substudy 1: Upadacitinib 30 mg vs Placebo; Test type: Superiority; p = 0.015, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Stratified by previous biologic use, baseline corticosteroid use and baseline Adapted Mayo score (≤ 7 and > 7); Adjusted risk difference (%) = 12.2, 95% CI 2-sided [2.3 to 22.0] — Difference = Upadacitinib 30 mg - Placebo
Statistical Analysis 4: Comparison: SS1: Placebo vs SS1: Upadacitinib 45 mg; Substudy 1: Upadacitinib 45 mg vs Placebo; Test type: Superiority; p = 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Stratified by previous biologic use, baseline corticosteroid use and baseline Adapted Mayo score (≤ 7 and > 7); Adjusted risk difference (%) = 20.1, 95% CI 2-sided [8.0 to 32.1] — Difference = Upadacitinib 45 mg - Placebo

6. Secondary Outcome: Substudy 1: Percentage Of Participants Achieving Clinical Response Per Adapted Mayo Score at Week 8
Description: The Adapted Mayo Score is a composite score of UC disease activity based on the following 3 subscores:
  1. Stool frequency subscore (SFS), scored from 0 (normal number of stools) to 3 (5 or more stools more than normal).
  2. Rectal bleeding subscore (RBS), scored from 0 (no blood seen) to 3 (blood alone passed).
  3. Endoscopic subscore, scored from 0 (normal or inactive disease) to 3 (severe disease, spontaneous bleeding, ulceration).
  The overall Adapted Mayo score ranges from 0 to 9 where higher scores represent more severe disease. Clinical response is defined as a decrease from baseline in the Adapted Mayo score ≥ 2 points and ≥ 30% from baseline, and a decrease in RBS ≥ 1 or an absolute RBS ≤ 1).
Time Frame: At Week 8
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | SS1: Placebo | SS1: Upadacitinib 7.5 mg | SS1: Upadacitinib 15 mg | SS1: Upadacitinib 30 mg | SS1: Upadacitinib 45 mg
Number analyzed (Participants) | 46 | 47 | 49 | 52 | 56
percentage of participants | 13.0 | 29.8 | 49.0 | 46.2 | 55.4
Statistical Analysis 1: Comparison: SS1: Placebo vs SS1: Upadacitinib 7.5 mg; Substudy 1: Upadacitinib 7.5 mg vs Placebo; Test type: Superiority; p = 0.038, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Stratified by previous biologic use, baseline corticosteroid use and baseline Adapted Mayo score (≤ 7 and > 7); Adjusted risk difference (%) = 16.7, 95% CI 2-sided [0.9 to 32.5] — Difference = Upadacitinib 7.5 mg - Placebo
Statistical Analysis 2: Comparison: SS1: Placebo vs SS1: Upadacitinib 15 mg; Substudy 1: Upadacitinib 15 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Stratified by previous biologic use, baseline corticosteroid use and baseline Adapted Mayo score (≤ 7 and > 7); Adjusted risk difference (%) = 35.2, 95% CI 2-sided [17.5 to 52.8] — Difference = Upadacitinib 15 mg - Placebo
Statistical Analysis 3: Comparison: SS1: Placebo vs SS1: Upadacitinib 30 mg; Substudy 1: Upadacitinib 30 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Stratified by previous biologic use, baseline corticosteroid use and baseline Adapted Mayo score (≤ 7 and > 7); Adjusted risk difference (%) = 33.6, 95% CI 2-sided [16.3 to 50.8] — Difference = Upadacitinib 30 mg - Placebo
Statistical Analysis 4: Comparison: SS1: Placebo vs SS1: Upadacitinib 45 mg; Substudy 1: Upadacitinib 45 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Stratified by previous biologic use, baseline corticosteroid use and baseline Adapted Mayo score (≤ 7 and > 7); Adjusted risk difference (%) = 45.1, 95% CI 2-sided [26.2 to 63.9] — Difference = Upadacitinib 45 mg - Placebo

7. Secondary Outcome: Substudy 1: Percentage Of Participants Achieving Clinical Response Per Partial Mayo Score at Week 2
Description: The Partial Mayo Score is a composite score of UC disease activity based on the following 2 subscores:
  1. Stool frequency subscore (SFS), scored from 0 (normal number of stools) to 3 (5 or more stools more than normal).
  2. Rectal bleeding subscore (RBS), scored from 0 (no blood seen) to 3 (blood alone passed).
  The overall Partial Mayo score ranges from 0 to 6 with higher scores representing more severe disease.
  Clinical response per Partial Mayo Score is defined as a decrease in Partial Adapted Mayo score ≥ 2 points and ≥ 30% from Baseline, plus a decrease in RBS ≥ 1 or an absolute RBS ≤ 1.
Time Frame: At Week 2
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | SS1: Placebo | SS1: Upadacitinib 7.5 mg | SS1: Upadacitinib 15 mg | SS1: Upadacitinib 30 mg | SS1: Upadacitinib 45 mg
Number analyzed (Participants) | 46 | 47 | 49 | 52 | 56
percentage of participants | 17.4 | 23.4 | 34.7 | 36.5 | 55.4
Statistical Analysis 1: Comparison: SS1: Placebo vs SS1: Upadacitinib 7.5 mg; Substudy 1: Upadacitinib 7.5 mg vs Placebo; Test type: Superiority; p = 0.495, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Stratified by previous biologic use, baseline corticosteroid use and baseline Adapted Mayo score (≤ 7 and > 7); Adjusted risk difference (%) = 5.9, 95% CI 2-sided [-11.1 to 22.9] — Difference = Upadacitinib 7.5 mg - Placebo
Statistical Analysis 2: Comparison: SS1: Placebo vs SS1: Upadacitinib 15 mg; Substudy 1: Upadacitinib 15 mg vs Placebo; Test type: Superiority; p = 0.074, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Stratified by previous biologic use, baseline corticosteroid use and baseline Adapted Mayo score (≤ 7 and > 7); Adjusted risk difference (%) = 15.9, 95% CI 2-sided [-1.6 to 33.4] — Difference = Upadacitinib 15 mg - Placebo
Statistical Analysis 3: Comparison: SS1: Placebo vs SS1: Upadacitinib 30 mg; Substudy 1: Upadacitinib 30 mg vs Placebo; Test type: Superiority; p = 0.033, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Stratified by previous biologic use, baseline corticosteroid use and baseline Adapted Mayo score (≤ 7 and > 7); Adjusted risk difference (%) = 19.2, 95% CI 2-sided [1.6 to 36.9] — Difference = Upadacitinib 30 mg - Placebo
Statistical Analysis 4: Comparison: SS1: Placebo vs SS1: Upadacitinib 45 mg; Substudy 1: Upadacitinib 45 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Stratified by previous biologic use, baseline corticosteroid use and baseline Adapted Mayo score (≤ 7 and > 7); Adjusted risk difference (%) = 40.1, 95% CI 2-sided [20.5 to 59.7] — Difference = Upadacitinib 45 mg - Placebo

8. Secondary Outcome: Substudy 1: Change in Full Mayo Score From Baseline to Week 8
Description: as for outcome 5
Time Frame: Baseline (Week 0), Week 8
Population: The Substudy 1 main population (ITT1A) includes participants who were randomized to at least one dose (placebo or upadacitinib 7.5 mg, 15 mg, 30 mg, 45 mg) during the main (initial) part of Substudy 1. Last observation carried forward (LOCF) was used for missing data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SS1: Placebo | SS1: Upadacitinib 7.5 mg | SS1: Upadacitinib 15 mg | SS1: Upadacitinib 30 mg | SS1: Upadacitinib 45 mg
Number analyzed (Participants) | 41 | 43 | 44 | 44 | 48
units on a scale | -0.741 (2.3302) | -2.870 (2.9685) | -3.589 (2.4984) | -4.211 (3.0886) | -4.606 (2.8976)
Statistical Analysis 1: Comparison: SS1: Placebo vs SS1: Upadacitinib 7.5 mg; Substudy 1: Upadacitinib 7.5 mg vs Placebo; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Stratified by previous biologic use, Baseline corticosteroid use, Baseline Adapted Mayo score (<= 7 and > 7)), and Baseline value as covariate; LS Mean Difference = -2.142, 95% CI 2-sided [-3.2323 to -1.0520] — Difference = Upadacitinib 7.5 mg - Placebo
Statistical Analysis 2: Comparison: SS1: Placebo vs SS1: Upadacitinib 15 mg; Substudy 1: Upadacitinib 15 mg vs Placebo; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 8, analysis 1]; LS Mean Difference = -2.938, 95% CI 2-sided [-4.0284 to -1.8478] — Difference = Upadacitinib 15 mg - Placebo
Statistical Analysis 3: Comparison: SS1: Placebo vs SS1: Upadacitinib 30 mg; Substudy 1: Upadacitinib 30 mg vs Placebo; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 8, analysis 1]; LS Mean Difference = -3.736, 95% CI 2-sided [-4.8247 to -2.6470] — Difference = Upadacitinib 30 mg - Placebo
Statistical Analysis 4: Comparison: SS1: Placebo vs SS1: Upadacitinib 45 mg; Substudy 1: Upadacitinib 45 mg vs Placebo; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 8, analysis 1]; LS Mean Difference = -4.061, 95% CI 2-sided [-5.1252 to -2.9974] — Difference = Upadacitinib 45 mg - Placebo

9. Secondary Outcome: Substudy 1: Percentage Of Participants With Endoscopic Remission at Week 8
Description: Endoscopic remission is defined as an endoscopic subscore of 0. Endoscopies were assessed by a blinded central reader and scored according to the following scale: 0 = Normal or inactive disease; 1 = Mild disease (erythema, decreased vascular pattern); 2 = Moderate disease (marked erythema, lack of vascular pattern, any friability, erosions); 3 = Severe disease (spontaneous bleeding, ulceration).
Time Frame: At Week 8
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | SS1: Placebo | SS1: Upadacitinib 7.5 mg | SS1: Upadacitinib 15 mg | SS1: Upadacitinib 30 mg | SS1: Upadacitinib 45 mg
Number analyzed (Participants) | 46 | 47 | 49 | 52 | 56
percentage of participants | 0 | 6.4 | 4.1 | 9.6 | 17.9
Statistical Analysis 1: Comparison: SS1: Placebo vs SS1: Upadacitinib 7.5 mg; Substudy 1: Upadacitinib 7.5 mg vs Placebo; Test type: Superiority; p = 0.075, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Stratified by previous biologic use, baseline corticosteroid use and baseline Adapted Mayo score (≤ 7 and > 7); Adjusted risk difference (%) = 6.6, 95% CI 2-sided [-0.7 to 13.9] — Difference = Upadacitinib 7.5 mg - Placebo
Statistical Analysis 2: Comparison: SS1: Placebo vs SS1: Upadacitinib 15 mg; Substudy 1: Upadacitinib 15 mg vs Placebo; Test type: Superiority; p = 0.199, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Stratified by previous biologic use, baseline corticosteroid use and baseline Adapted Mayo score (≤ 7 and > 7); Adjusted risk difference (%) = 3.8, 95% CI 2-sided [-2.0 to 9.6] — Difference = Upadacitinib 15 mg - Placebo
Statistical Analysis 3: Comparison: SS1: Placebo vs SS1: Upadacitinib 30 mg; Substudy 1: Upadacitinib 30 mg vs Placebo; Test type: Superiority; p = 0.015, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Stratified by previous biologic use, baseline corticosteroid use and baseline Adapted Mayo score (≤ 7 and > 7); Adjusted risk difference (%) = 11.1, 95% CI 2-sided [2.2 to 20.0] — Difference = Upadacitinib 30 mg - Placebo
Statistical Analysis 4: Comparison: SS1: Placebo vs SS1: Upadacitinib 45 mg; Substudy 1: Upadacitinib 45 mg vs Placebo; Test type: Superiority; p = 0.004, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Stratified by previous biologic use, baseline corticosteroid use and baseline Adapted Mayo score (≤ 7 and > 7); Adjusted risk difference (%) = 17.8, 95% CI 2-sided [5.8 to 29.9] — Difference = Upadacitinib 45 mg - Placebo

10. Secondary Outcome: Substudy 1: Percentage Of Participants Who Achieved Histologic Improvement at Week 8
Description: The Geboes histologic index includes seven histological features (architectural change, chronic inflammatory infiltrate, lamina propria neutrophils and eosinophils, neutrophils in epithelium, crypt destruction and erosion or ulcers). The Geboes score has 6 grades, each with 3-5 subgrades: Grade 0, structural change only; Grade 1, chronic inflammation; Grade 2, lamina propria neutrophils and eosinophils; Grade 3, neutrophils in epithelium; Grade 4, crypt destruction; and Grade 5, erosions or ulceration.
  Histologic improvement was defined as decrease from baseline in Geboes score.
Time Frame: At Week 8
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | SS1: Placebo | SS1: Upadacitinib 7.5 mg | SS1: Upadacitinib 15 mg | SS1: Upadacitinib 30 mg | SS1: Upadacitinib 45 mg
Number analyzed (Participants) | 46 | 47 | 49 | 52 | 56
percentage of participants | 6.5 | 31.9 | 51.0 | 44.2 | 48.2
Statistical Analysis 1: Comparison: SS1: Placebo vs SS1: Upadacitinib 7.5 mg; Substudy 1: Upadacitinib 7.5 mg vs Placebo; Test type: Superiority; p = 0.003, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Stratified by previous biologic use, baseline corticosteroid use and baseline Adapted Mayo score (≤ 7 and > 7); Adjusted risk difference (%) = 25.6, 95% CI 2-sided [8.9 to 42.3] — Difference = Upadacitinib 7.5 mg - Placebo
Statistical Analysis 2: Comparison: SS1: Placebo vs SS1: Upadacitinib 15 mg; Substudy 1: Upadacitinib 15 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Stratified by previous biologic use, baseline corticosteroid use and baseline Adapted Mayo score (≤ 7 and > 7); Adjusted risk difference (%) = 43.6, 95% CI 2-sided [25.4 to 61.8] — Difference = Upadacitinib 15 mg - Placebo
Statistical Analysis 3: Comparison: SS1: Placebo vs SS1: Upadacitinib 30 mg; Substudy 1: Upadacitinib 30 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Stratified by previous biologic use, baseline corticosteroid use and baseline Adapted Mayo score (≤ 7 and > 7); Adjusted risk difference (%) = 39.4, 95% CI 2-sided [21.3 to 57.5] — Difference = Upadacitinib 30 mg - Placebo
Statistical Analysis 4: Comparison: SS1: Placebo vs SS1: Upadacitinib 45 mg; Substudy 1: Upadacitinib 45 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Stratified by previous biologic use, baseline corticosteroid use and baseline Adapted Mayo score (≤ 7 and > 7); Adjusted risk difference (%) = 43.1, 95% CI 2-sided [24.4 to 61.9] — Difference = Upadacitinib 45 mg - Placebo

11. Secondary Outcome: Substudy 2: Percentage Of Participants With Endoscopic Improvement at Week 8
Description: as for outcome 4
Time Frame: At Week 8
Population: The Substudy 2, Part 1 population (ITT1) includes all randomized participants in the 8-week double-blind induction period who received at least one dose of double-blinded study drug in Part 1; NRI incorporating multiple imputation (MI) to handle missing data due to COVID-19 (NRI-C) was used with participants analyzed according to treatment groups to which they were randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SS2: Placebo | SS2: Upadacitinib 45 mg
Number analyzed (Participants) | 154 | 319
percentage of participants | 7.4 [3.2 to 11.5] | 36.3 [31.0 to 41.7]
Statistical Analysis 1: Comparison: SS2: Placebo vs SS2: Upadacitinib 45 mg; Substudy 2: Upadacitinib 45 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Stratified by bio-IR status (bio-IR vs. non-bio-IR), Baseline corticosteroid use (yes or no) and Baseline Adapted Mayo score (≤ 7 vs. > 7); Adjusted risk difference (%) = 29.3, 95% CI 2-sided [22.6 to 35.9] — Difference = Upadacitinib 45 mg - Placebo

12. Secondary Outcome: Substudy 2: Percentage Of Participants With Endoscopic Remission at Week 8
Description: as for outcome 9
Time Frame: At Week 8
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SS2: Placebo | SS2: Upadacitinib 45 mg
Number analyzed (Participants) | 154 | 319
percentage of participants | 1.3 [0.0 to 3.1] | 13.7 [9.9 to 17.6]
Statistical Analysis 1: Comparison: SS2: Placebo vs SS2: Upadacitinib 45 mg; Substudy 2: Upadacitinib 45 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 11, analysis 1]; Adjusted risk difference (%) = 12.7, 95% CI 2-sided [8.4 to 17.0] — Difference = Upadacitinib 45 mg - Placebo

13. Secondary Outcome: Substudy 2: Percentage Of Participants Achieving Clinical Response Per Adapted Mayo Score at Week 8
Description: as for outcome 6
Time Frame: At Week 8
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SS2: Placebo | SS2: Upadacitinib 45 mg
Number analyzed (Participants) | 154 | 319
percentage of participants | 27.3 [20.2 to 34.3] | 72.6 [67.7 to 77.5]
Statistical Analysis 1: Comparison: SS2: Placebo vs SS2: Upadacitinib 45 mg; Substudy 2: Upadacitinib 45 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 11, analysis 1]; Adjusted risk difference (%) = 46.3, 95% CI 2-sided [38.4 to 54.2] — Difference = Upadacitinib 45 mg - Placebo

14. Secondary Outcome: Substudy 2: Percentage Of Participants Achieving Clinical Response Per Partial Mayo Score at Week 2
Description: The Partial Mayo Score is a composite score of UC disease activity based on the following 2 subscores:
  1. Stool frequency subscore (SFS), scored from 0 (normal number of stools) to 3 (5 or more stools more than normal).
  2. Rectal bleeding subscore (RBS), scored from 0 (no blood seen) to 3 (blood alone passed).
  The overall Partial Mayo score ranges from 0 to 6 with higher scores representing more severe disease.
  Clinical response per Partial Mayo Score is defined as a decrease from Baseline ≥ 1 point and ≥ 30% from Baseline, plus a decrease in RBS ≥ 1 or an absolute RBS ≤ 1.
Time Frame: At Week 2
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SS2: Placebo | SS2: Upadacitinib 45 mg
Number analyzed (Participants) | 154 | 319
percentage of participants | 27.3 [20.2 to 34.3] | 60.1 [54.7 to 65.5]
Statistical Analysis 1: Comparison: SS2: Placebo vs SS2: Upadacitinib 45 mg; Substudy 2: Upadacitinib 45 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 11, analysis 1]; Adjusted risk difference (%) = 33.3, 95% CI 2-sided [24.8 to 41.8]; Difference = Upadacitinib 45 mg - Placebo

15. Secondary Outcome: Substudy 2: Percentage Of Participants Who Achieved Histologic-Endoscopic Mucosal Improvement at Week 8
Description: Histologic-endoscopic mucosal improvement is defined as an endoscopic subscore of 0 or 1 and a Geboes score ≤ 3.1.
  The endoscopic subscore ranges from 0 (normal or inactive disease) to 3 (severe disease with spontaneous bleeding, ulceration).
  The Geboes histologic index includes seven histological features (architectural change, chronic inflammatory infiltrate, lamina propria neutrophils and eosinophils, neutrophils in epithelium, crypt destruction and erosion or ulcers). The Geboes score has 6 grades, each with 3-5 subgrades: Grade 0, structural change only; Grade 1, chronic inflammation; Grade 2, lamina propria neutrophils and eosinophils; Grade 3, neutrophils in epithelium; Grade 4, crypt destruction; and Grade 5, erosions or ulceration.
Time Frame: At Week 8
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SS2: Placebo | SS2: Upadacitinib 45 mg
Number analyzed (Participants) | 154 | 319
percentage of participants | 6.6 [2.6 to 10.5] | 30.1 [25.0 to 35.1]
Statistical Analysis 1: Comparison: SS2: Placebo vs SS2: Upadacitinib 45 mg; Substudy 2: Upadacitinib 45 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 11, analysis 1]; Adjusted risk difference (%) = 23.7, 95% CI 2-sided [17.5 to 30.0] — Difference = Upadacitinib 45 mg - Placebo

16. Secondary Outcome: Substudy 2: Percentage Of Participants Who Report No Bowel Urgency at Week 8
Description: Bowel urgency was assessed by participants in a subject diary completed once a day.
Time Frame: At Week 8
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SS2: Placebo | SS2: Upadacitinib 45 mg
Number analyzed (Participants) | 154 | 319
percentage of participants | 21.4 [14.9 to 27.9] | 48.4 [42.9 to 53.9]
Statistical Analysis 1: Comparison: SS2: Placebo vs SS2: Upadacitinib 45 mg; Substudy 2: Upadacitinib 45 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 11, analysis 1]; Adjusted risk difference (%) = 27.4, 95% CI 2-sided [19.2 to 35.6] — Difference = Upadacitinib 45 mg - Placebo

17. Secondary Outcome: Substudy 2: Percentage Of Participants Who Reported No Abdominal Pain at Week 8
Description: Abdominal pain was assessed by participants in a subject diary completed once a day.
Time Frame: At Week 8
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SS2: Placebo | SS2: Upadacitinib 45 mg
Number analyzed (Participants) | 154 | 319
percentage of participants | 23.4 [16.7 to 30.1] | 46.6 [41.1 to 52.1]
Statistical Analysis 1: Comparison: SS2: Placebo vs SS2: Upadacitinib 45 mg; Substudy 2: Upadacitinib 45 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 11, analysis 1]; Adjusted risk difference (%) = 23.6, 95% CI 2-sided [15.1 to 32.1] — Difference = Upadacitinib 45 mg - Placebo

18. Secondary Outcome: Substudy 2: Percentage Of Participants Who Achieved Histologic Improvement at Week 8
Description: as for outcome 10
Time Frame: At Week 8
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SS2: Placebo | SS2: Upadacitinib 45 mg
Number analyzed (Participants) | 154 | 319
percentage of participants | 22.5 [15.9 to 29.1] | 55.0 [49.5 to 60.5]
Statistical Analysis 1: Comparison: SS2: Placebo vs SS2: Upadacitinib 45 mg; Substudy 2: Upadacitinib 45 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 11, analysis 1]; Adjusted risk difference (%) = 32.2, 95% CI 2-sided [23.8 to 40.7] — Difference = Upadacitinib 45 mg - Placebo

19. Secondary Outcome: Substudy 2: Change From Baseline in Inflammatory Bowel Disease Questionnaire (IBDQ) Total Score at Week 8
Description: The Inflammatory Bowel Disease Questionnaire (IBDQ) is used to assess health-related quality of life (HRQoL) in patients with ulcerative colitis. It consists of 32 questions evaluating bowel and systemic symptoms, as well as emotional and social functions. Each question is answered on a scale from 1 (worst) to 7 (best). The total score ranges from 32 to 224 with higher scores indicating better health-related quality of life. A positive change from Baseline indicates improvement.
Time Frame: Baseline (Week 0), Week 8
Population: The Substudy 2, Part 1 ITT1 population with available data; a mixed effect model repeat measurement (MMRM) analysis with data from observed cases up to Week 8 was used except for measurements at or after the occurrence of UC-related corticosteroids intercurrent event were excluded
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | SS2: Placebo | SS2: Upadacitinib 45 mg
Number analyzed (Participants) | 125 | 292
units on a scale | 21.7 [16.03 to 27.28] | 55.3 [51.54 to 59.15]
Statistical Analysis 1: Comparison: SS2: Placebo vs SS2: Upadacitinib 45 mg; Substudy 2: Upadacitinib 45 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed-effect model repeated measurement — [p-value comment as in outcome 1, analysis 1]; MMRM with Baseline, treatment, visit, treatment-by-visit interaction, and strata (Baseline Adapted Mayo score, corticosteroid use, and bio-IR status); Least Squares (LS) Mean Difference = 33.7, 95% CI 2-sided [27.02 to 40.36], Standard Error of Mean 3.39 — Difference = Upadacitinib 45 mg - Placebo

20. Secondary Outcome: Substudy 2: Percentage Of Participants With Mucosal Healing at Week 8
Description: Mucosal healing is defined as an endoscopic score of 0 and Geboes score < 2.0. The endoscopic subscore ranges from 0 (normal or inactive disease) to 3 (severe disease with spontaneous bleeding, ulceration).
  The Geboes histologic index includes seven histological features (architectural change, chronic inflammatory infiltrate, lamina propria neutrophils and eosinophils, neutrophils in epithelium, crypt destruction and erosion or ulcers). The Geboes score has 6 grades, each with 3-5 subgrades: Grade 0, structural change only; Grade 1, chronic inflammation; Grade 2, lamina propria neutrophils and eosinophils; Grade 3, neutrophils in epithelium; Grade 4, crypt destruction; and Grade 5, erosions or ulceration.
Time Frame: At Week 8
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SS2: Placebo | SS2: Upadacitinib 45 mg
Number analyzed (Participants) | 154 | 319
percentage of participants | 1.3 [0.0 to 3.1] | 10.7 [7.3 to 14.1]
Statistical Analysis 1: Comparison: SS2: Placebo vs SS2: Upadacitinib 45 mg; Substudy 2: Upadacitinib 45 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Stratified by Baseline corticosteroid use (yes or no), Baseline Adapted Mayo score (≤ 7 or > 7), and bio-IR status (bio-IR or non-bio-IR); Adjusted risk difference (%) = 9.7, 95% CI 2-sided [5.7 to 13.7] — Difference = Upadacitinib 45 mg - Placebo

21. Secondary Outcome: Substudy 2: Change From Baseline in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Score at Week 8
Description: The FACIT fatigue questionnaire was developed to assess fatigue associated with anemia. It consists of 13 fatigue-related questions. Each question is answered on a 5-point Likert scale: 0 (not at all); 1 (a little bit); 2 (somewhat); 3 (quite a bit); and 4 (very much). The total score ranges from 0 to 52, where higher scores represent less fatigue, and a positive change from Baseline indicates improvement.
Time Frame: Baseline (Week 0), Week 8
Population: as for outcome 19
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | SS2: Placebo | SS2: Upadacitinib 45 mg
Number analyzed (Participants) | 125 | 291
units on a scale | 2.8 [1.23 to 4.44] | 9.5 [8.44 to 10.61]
Statistical Analysis 1: Comparison: SS2: Placebo vs SS2: Upadacitinib 45 mg; Substudy 2: Upadacitinib 45 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed-effect model repeated measurement — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 19, analysis 1]; Least Squares (LS) Mean Difference = 6.7, 95% CI 2-sided [4.79 to 8.59], Standard Error of Mean 0.97 — Difference = Upadacitinib 45 mg - Placebo

22. Secondary Outcome: Substudy 3: Percentage Of Participants With Endoscopic Improvement at Week 52
Description: as for outcome 4
Time Frame: At Week 52
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SS3: Placebo | SS3: UPA 15 mg | SS3: UPA 30 mg
Number analyzed (Participants) | 149 | 148 | 154
percentage of participants | 14.5 [8.7 to 20.3] | 48.7 [40.5 to 56.8] | 61.6 [53.6 to 69.6]
Statistical Analysis 1: Comparison: SS3: Placebo vs SS3: UPA 15 mg; Substudy 3: Upadacitinib 15 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — The primary and ranked secondary efficacy endpoints were tested with graphical multiplicity adjustment to ensure a strong control of family-wise type I error rate at significance level α= 0.05 (2-sided); Stratified by Bio-IR (Bio-IR/Non-Bio-IR) at Induction Study Baseline; clinical remission at Week 0 (yes/no); corticosteroid use at Week 0 (yes/no); Adjusted risk difference (%) = 34.4, 95% CI 2-sided [25.1 to 43.7] — Difference = Upadacitinib 15 mg - Placebo
Statistical Analysis 2: Comparison: SS3: Placebo vs SS3: UPA 30 mg; Substudy 3: Upadacitinib 30 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 22, analysis 1]; [statistical method as in outcome 22, analysis 1]; Adjusted risk difference (%) = 46.3, 95% CI 2-sided [36.7 to 55.8] — Difference = Upadacitinib 30 mg - Placebo

23. Secondary Outcome: Substudy 3: Percentage of Participants With Clinical Remission Per Adapted Mayo Score at Week 52 Among Those Who Achieved Clinical Remission at the End of the Induction Treatment
Description: as for outcome 3
Time Frame: At Week 52
Population: Substudy 3 ITT_A population: the first 451 upadacitinib 45 mg 8-week induction responders who were enrolled under the protocol for 52-week maintenance treatment period in Cohort 1 and who achieved clinical remission per Adapted Mayo Score in Substudy 1, 2, or M14-675. Non-responder imputation incorporating multiple imputation (MI) to handle missing data due to COVID-19 (NRI-C) was used to handle missing data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SS3: Placebo | SS3: UPA 15 mg | SS3: UPA 30 mg
Number analyzed (Participants) | 54 | 47 | 58
percentage of participants | 22.2 [11.1 to 33.3] | 59.2 [45.1 to 73.4] | 69.7 [57.7 to 81.8]
Statistical Analysis 1: Comparison: SS3: Placebo vs SS3: UPA 15 mg; Substudy 3: Upadacitinib 15 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 22, analysis 1]; [statistical method as in outcome 22, analysis 1]; Adjusted risk difference (%) = 37.4, 95% CI 2-sided [20.3 to 54.6] — Difference = Upadacitinib 15 mg - Placebo
Statistical Analysis 2: Comparison: SS3: Placebo vs SS3: UPA 30 mg; Substudy 3: Upadacitinib 30 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 22, analysis 1]; [statistical method as in outcome 22, analysis 1]; Adjusted risk difference (%) = 47.0, 95% CI 2-sided [30.7 to 63.3] — Difference = Upadacitinib 30 mg - Placebo

24. Secondary Outcome: Substudy 3: Percentage of Participants Who Achieved Clinical Remission Per Adapted Mayo Score at Wk 52 and Were Corticosteroid Free for ≥ 90 Days Immediately Preceding Wk 52 Among Those Who Achieved Clinical Remission at the End of the Induction Treatment
Description: as for outcome 3
Time Frame: At Week 52
Population: as for outcome 23
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- SS3: Placebo: Participants who achieved clinical response in Substudy 1, Substudy 2, or Study M14-675 at Week 8, while receiving upadacitinib 15, 30, or 45 mg QD and were randomized to placebo QD in Substudy 3 for up to 52 weeks. In addition, participants who received double-blind placebo QD treatment for 8 weeks during Substudy1, Substudy 2 Part 1, or Study M14-675 Part 1 and achieved clinical response at Week 8 continued to receive blinded placebo QD in Substudy 3 for up to 52 weeks.
Arm/Group | SS3: Placebo | SS3: UPA 15 mg | SS3: UPA 30 mg
Number analyzed (Participants) | 54 | 47 | 58
percentage of participants | 22.2 [11.1 to 33.3] | 57.1 [42.9 to 71.3] | 68.0 [55.8 to 80.2]
Statistical Analysis 1: Comparison: SS3: Placebo vs SS3: UPA 15 mg; Substudy 3: Upadacitinib 15 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 22, analysis 1]; [statistical method as in outcome 22, analysis 1]; Adjusted risk difference (%) = 35.4, 95% CI 2-sided [18.2 to 52.7] — Difference = Upadacitinib 15 mg - Placebo
Statistical Analysis 2: Comparison: SS3: Placebo vs SS3: UPA 30 mg; Substudy 3: Upadacitinib 30 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 22, analysis 1]; [statistical method as in outcome 22, analysis 1]; Adjusted risk difference (%) = 45.1, 95% CI 2-sided [28.7 to 61.6] — Difference = Upadacitinib 30 mg - Placebo

25. Secondary Outcome: Substudy 3: Percentage of Participants With Endoscopic Improvement at Wk 52 Among Those Who Achieved Endoscopic Improvement at the End of the Induction Treatment
Description: as for outcome 4
Time Frame: At Week 52
Population: Substudy 3 ITT_A population: the first 451 upadacitinib 45 mg 8-week induction responders who were enrolled under the protocol for 52-week maintenance treatment period in Cohort 1 and who achieved endoscopic improvement in Substudy 1, 2, or M14-675. Non-responder imputation incorporating multiple imputation (MI) to handle missing data due to COVID-19 (NRI-C) was used to handle missing data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SS3: Placebo | SS3: UPA 15 mg | SS3: UPA 30 mg
Number analyzed (Participants) | 73 | 63 | 79
percentage of participants | 19.2 [9.9 to 28.4] | 61.6 [49.6 to 73.7] | 69.5 [59.1 to 80.0]
Statistical Analysis 1: Comparison: SS3: Placebo vs SS3: UPA 15 mg; Substudy 3: Upadacitinib 15 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 22, analysis 1]; [statistical method as in outcome 22, analysis 1]; Adjusted risk difference (%) = 42.0, 95% CI 2-sided [27.8 to 56.2] — Difference = Upadacitinib 15 mg - Placebo
Statistical Analysis 2: Comparison: SS3: Placebo vs SS3: UPA 30 mg; Substudy 3: Upadacitinib 30 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 22, analysis 1]; [statistical method as in outcome 22, analysis 1]; Adjusted risk difference (%) = 48.6, 95% CI 2-sided [35.5 to 61.7] — Difference = Upadacitinib 30 mg - Placebo

26. Secondary Outcome: Substudy 3: Percentage Of Participants With Endoscopic Remission At Week 52
Description: as for outcome 9
Time Frame: At Week 52
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SS3: Placebo | SS3: UPA 15 mg | SS3: UPA 30 mg
Number analyzed (Participants) | 149 | 148 | 154
percentage of participants | 5.6 [1.8 to 9.3] | 24.2 [17.3 to 31.2] | 25.9 [18.8 to 33.0]
Statistical Analysis 1: Comparison: SS3: Placebo vs SS3: UPA 15 mg; Substudy 3: Upadacitinib 15 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 22, analysis 1]; [statistical method as in outcome 22, analysis 1]; Adjusted risk difference (%) = 18.7, 95% CI 2-sided [11.0 to 26.4] — Difference = Upadacitinib 15 mg - Placebo
Statistical Analysis 2: Comparison: SS3: Placebo vs SS3: UPA 30 mg; Substudy 3: Upadacitinib 30 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 22, analysis 1]; [statistical method as in outcome 22, analysis 1]; Adjusted risk difference (%) = 19.4, 95% CI 2-sided [11.7 to 27.2] — Difference = Upadacitinib 30 mg - Placebo

27. Secondary Outcome: Substudy 3: Percentage Of Participants Who Maintained Clinical Response Per Adapted Mayo Score at Wk 52 Among Those Who Achieved Clinical Response at the End of the Induction Treatment
Description: as for outcome 6
Time Frame: At Week 52
Population: Substudy 3 ITT_A population: the first 451 upadacitinib 45 mg 8-week induction responders who were enrolled under the protocol for 52-week maintenance treatment period in Cohort 1 and who achieved clinical response per Adapted Mayo Score in Substudy 1, 2, or M14-675. Non-responder imputation incorporating multiple imputation (MI) to handle missing data due to COVID-19 (NRI-C) was used to handle missing data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SS3: Placebo | SS3: UPA 15 mg | SS3: UPA 30 mg
Number analyzed (Participants) | 134 | 135 | 144
percentage of participants | 18.8 [12.1 to 25.5] | 63.0 [54.8 to 71.1] | 76.6 [69.6 to 83.6]
Statistical Analysis 1: Comparison: SS3: Placebo vs SS3: UPA 15 mg; Substudy 3: Upadacitinib 15 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 22, analysis 1]; [statistical method as in outcome 22, analysis 1]; Adjusted risk difference (%) = 44.6, 95% CI 2-sided [34.5 to 54.7] — Difference = Upadacitinib 15 mg - Placebo
Statistical Analysis 2: Comparison: SS3: Placebo vs SS3: UPA 30 mg; Substudy 3: Upadacitinib 30 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 22, analysis 1]; [statistical method as in outcome 22, analysis 1]; Adjusted risk difference (%) = 56.6, 95% CI 2-sided [47.2 to 66.0] — Difference = Upadacitinib 30 mg - Placebo

28. Secondary Outcome: Substudy 3: Percentage Of Participants Who Achieved Histologic-Endoscopic Mucosal Improvement at Week 52
Description: as for outcome 15
Time Frame: At Week 52
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SS3: Placebo | SS3: UPA 15 mg | SS3: UPA 30 mg
Number analyzed (Participants) | 149 | 148 | 154
percentage of participants | 11.9 [6.7 to 17.2] | 35.0 [27.1 to 42.8] | 49.8 [41.5 to 58.0]
Statistical Analysis 1: Comparison: SS3: Placebo vs SS3: UPA 15 mg; Substudy 3: Upadacitinib 15 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 22, analysis 1]; [statistical method as in outcome 22, analysis 1]; Adjusted risk difference (%) = 23.8, 95% CI 2-sided [14.8 to 32.8] — Difference = Upadacitinib 15 mg - Placebo
Statistical Analysis 2: Comparison: SS3: Placebo vs SS3: UPA 30 mg; Substudy 3: Upadacitinib 30 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 22, analysis 1]; [statistical method as in outcome 22, analysis 1]; Adjusted risk difference (%) = 37.3, 95% CI 2-sided [27.8 to 46.8] — Difference = Upadacitinib 30 mg - Placebo

29. Secondary Outcome: Substudy 3: Change From Baseline in Inflammatory Bowel Disease Questionnaire (IBDQ) Total Score at Week 52
Description: as for outcome 19
Time Frame: Baseline (Week 0), Week 52
Population: Substudy 3 ITT_A population with available data: Baseline is defined as the last non-missing value prior to the first dose in Phase 2b Induction or Induction Studies. Multiple Imputation Incorporating Return-to-Baseline (RTB-MI) was used to handle missing data.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | SS3: Placebo | SS3: UPA 15 mg | SS3: UPA 30 mg
Number analyzed (Participants) | 149 | 148 | 154
units on a scale | 17.9 [10.79 to 25.00] | 49.2 [42.59 to 55.89] | 58.9 [52.14 to 65.59]
Statistical Analysis 1: Comparison: SS3: Placebo vs SS3: UPA 15 mg; Substudy 3: Upadacitinib 15 mg vs Placebo; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 22, analysis 1]; Stratified by corticosteroid use at Week 0 (yes/no); clinical remission status at Week 0 (yes/ no); Bio-IR status at Baseline (Bio-IR or Non-Bio-IR); LS Mean Difference = 31.3, 95% CI 2-sided [21.98 to 40.70], Standard Error of Mean 4.77 — Difference = Upadacitinib 15 mg - Placebo
Statistical Analysis 2: Comparison: SS3: Placebo vs SS3: UPA 30 mg; Substudy 3: Upadacitinib 30 mg vs Placebo; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 22, analysis 1]; [statistical method as in outcome 29, analysis 1]; LS Mean Difference = 41.0, 95% CI 2-sided [31.39 to 50.55], Standard Error of Mean 4.88 — Difference = Upadacitinib 30 mg - Placebo

30. Secondary Outcome: Substudy 3: Percentage Of Participants With Mucosal Healing at Week 52
Description: as for outcome 20
Time Frame: At Week 52
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SS3: Placebo | SS3: UPA 15 mg | SS3: UPA 30 mg
Number analyzed (Participants) | 149 | 148 | 154
percentage of participants | 4.7 [1.3 to 8.2] | 17.6 [11.4 to 23.8] | 19.0 [12.6 to 25.4]
Statistical Analysis 1: Comparison: SS3: Placebo vs SS3: UPA 15 mg; Substudy 3: Upadacitinib 15 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 22, analysis 1]; [statistical method as in outcome 22, analysis 1]; Adjusted risk difference (%) = 13.0, 95% CI 2-sided [6.0 to 20.0] — Difference = Upadacitinib 15 mg - Placebo
Statistical Analysis 2: Comparison: SS3: Placebo vs SS3: UPA 30 mg; Substudy 3: Upadacitinib 30 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 22, analysis 1]; [statistical method as in outcome 22, analysis 1]; Adjusted risk difference (%) = 13.6, 95% CI 2-sided [6.6 to 20.6] — Difference = Upadacitinib 30 mg - Placebo

31. Secondary Outcome: Substudy 3: Percentage Of Participants Who Reported No Bowel Urgency at Week 52
Description: Bowel urgency was assessed by participants in a subject diary completed once a day.
Time Frame: At Week 52
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SS3: Placebo | SS3: UPA 15 mg | SS3: UPA 30 mg
Number analyzed (Participants) | 149 | 148 | 154
percentage of participants | 17.4 [11.4 to 23.5] | 56.1 [48.1 to 64.1] | 63.6 [56.0 to 71.2]
Statistical Analysis 1: Comparison: SS3: Placebo vs SS3: UPA 15 mg; Substudy 3: Upadacitinib 15 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 22, analysis 1]; [statistical method as in outcome 22, analysis 1]; Adjusted risk difference (%) = 38.7, 95% CI 2-sided [28.9 to 48.5] — Difference = Upadacitinib 15 mg - Placebo
Statistical Analysis 2: Comparison: SS3: Placebo vs SS3: UPA 30 mg; Substudy 3: Upadacitinib 30 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 22, analysis 1]; [statistical method as in outcome 22, analysis 1]; Adjusted risk difference (%) = 45.1, 95% CI 2-sided [35.5 to 54.8] — Difference = Upadacitinib 30 mg - Placebo

32. Secondary Outcome: Substudy 3: Percentage Of Participants Who Reported No Abdominal Pain at Week 52
Description: Abdominal pain was assessed by participants in a subject diary completed once a day.
Time Frame: At Week 52
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SS3: Placebo | SS3: UPA 15 mg | SS3: UPA 30 mg
Number analyzed (Participants) | 149 | 148 | 154
percentage of participants | 20.8 [14.2 to 27.3] | 45.9 [37.9 to 54.0] | 55.3 [47.4 to 63.2]
Statistical Analysis 1: Comparison: SS3: Placebo vs SS3: UPA 15 mg; Substudy 3: Upadacitinib 15 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 22, analysis 1]; [statistical method as in outcome 22, analysis 1]; Adjusted risk difference (%) = 24.3, 95% CI 2-sided [14.2 to 34.5] — Difference = Upadacitinib 15 mg - Placebo
Statistical Analysis 2: Comparison: SS3: Placebo vs SS3: UPA 30 mg; Substudy 3: Upadacitinib 30 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 22, analysis 1]; [statistical method as in outcome 22, analysis 1]; Adjusted risk difference (%) = 33.7, 95% CI 2-sided [23.6 to 43.9] — Difference = Upadacitinib 30 mg - Placebo

33. Secondary Outcome: Substudy 3: Change From Baseline in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Score at Week 52
Description: as for outcome 21
Time Frame: Baseline (Week 0), Week 52
Population: as for outcome 29
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | SS3: Placebo | SS3: UPA 15 mg | SS3: UPA 30 mg
Number analyzed (Participants) | 149 | 148 | 154
units on a scale | 3.7 [1.88 to 5.43] | 8.7 [7.01 to 10.49] | 9.5 [7.80 to 11.22]
Statistical Analysis 1: Comparison: SS3: Placebo vs SS3: UPA 15 mg; Substudy 3: Upadacitinib 15 mg vs Placebo; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 22, analysis 1]; Stratified by corticosteroid use at Week 0 (yes/no); clinical remission status at Week 0 (yes/no); Bio-IR status at Baseline (Bio-IR or Non-Bio-IR); LS Mean Difference = 5.1, 95% CI 2-sided [2.67 to 7.52] — Difference = Upadacitinib 15 mg - Placebo
Statistical Analysis 2: Comparison: SS3: Placebo vs SS3: UPA 30 mg; Substudy 3: Upadacitinib 30 mg vs Placebo; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 22, analysis 1]; [statistical method as in outcome 33, analysis 1]; LS Mean Difference = 5.9, 95% CI 2-sided [3.44 to 8.27] — Difference = Upadacitinib 30 mg - Placebo

ADVERSE EVENTS:
Time Frame: All-cause mortality is reported from enrollment to end of study; median time on follow-up was up to 57, 61, and 364 days for Substudies 1, 2, and 3, respectively. TEAEs and SAEs were collected from first dose of study drug until 30 days after last dose of study drug; mean duration on study drug was up to 57, 56, and 364 days for Substudies 1, 2, and 3, respectively.
Description: For safety analyses, participants were assigned to a treatment group based on the treatment actually received, regardless of the treatment randomized. The "as treated" group was determined by the most frequent dose regimen received in the analysis period.
Groups:
- SS3: Upadacitinib 7.5 mg: Participants who received double-blinded treatment of upadacitinib 7.5 mg QD for 8 weeks during Substudy 1 and achieved clinical response at Week 8 continued to receive blinded treatment of upadacitinib 7.5 mg QD in Substudy 3 for up to 52 weeks.
- SS3: Upadacitinib 15 mg: Participants who achieved clinical response in Substudy 1, Substudy 2, or Study M14-675 at either Week 8 or Week 16, while receiving upadacitinib 15, 30, or 45 mg QD and those who achieved clinical response while receiving upadacitinib 15 mg QD in Substudy 1 and were randomized to upadacitinib 15 mg QD in Substudy 3 for up to 52 weeks. In addition, participants who received upadacitinib 45 mg QD in Induction Phase and did not achieve clinical response and received upadacitinib 45 mg QD in Extended Treatment in Substudy 2 Part 2 or in Study M14-675 Part 2 and achieved clinical response at Week 16 and were randomized to upadacitinib 15 mg QD in Substudy 3.
- SS3: Upadacitinib 30 mg: Participants who achieved clinical response in Substudy 1, Substudy 2, or Study M14-675 at either Week 8 or Week 16, while receiving upadacitinib 15, 30, or 45 mg QD and those who achieved clinical response while receiving upadacitinib 15 mg QD in Substudy 1 and were randomized to upadacitinib 30 mg QD in Substudy 3 for up to 52 weeks. In addition, participants who received upadacitinib 45 mg QD in Induction Phase and did not achieve clinical response and received upadacitinib 45 mg QD in Extended Treatment in Substudy 2 Part 2 or in Study M14-675 Part 2 and achieved clinical response at Week 16 and were randomized to upadacitinib 30 mg QD in Substudy 3.
Arm/Group | SS1: Placebo | SS1: Upadacitinib 7.5 mg | SS1: Upadacitinib 15 mg | SS1: Upadacitinib 30 mg | SS1: Upadacitinib 45 mg | SS2: Placebo | SS2: Upadacitinib 45 mg | SS2: Placebo/Upadacitinib 45 mg | SS2: Upadacitinib 45 mg/Upadacitinib 45 mg | SS3: Placebo | SS3: Upadacitinib 7.5 mg | SS3: Upadacitinib 15 mg | SS3: Upadacitinib 30 mg
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/47 | 0/49 | 0/117 | 0/123 | 0/155 | 0/319 | 0/85 | 0/59 | 0/385 | 0/20 | 0/323 | 0/316
Serious Adverse Events (participants affected / at risk) | 5/46 | 0/47 | 2/49 | 5/117 | 6/123 | 9/155 | 8/319 | 2/85 | 2/59 | 32/385 | 0/20 | 24/323 | 25/316
Other Adverse Events (participants affected / at risk) | 27/46 | 18/47 | 22/49 | 58/117 | 50/123 | 62/155 | 121/319 | 36/85 | 17/59 | 216/385 | 18/20 | 181/323 | 166/316
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SS1: Placebo (N=46) | SS1: Upadacitinib 7.5 mg (N=47) | SS1: Upadacitinib 15 mg (N=49) | SS1: Upadacitinib 30 mg (N=117) | SS1: Upadacitinib 45 mg (N=123) | SS2: Placebo (N=155) | SS2: Upadacitinib 45 mg (N=319) | SS2: Placebo/Upadacitinib 45 mg (N=85) | SS2: Upadacitinib 45 mg/Upadacitinib 45 mg (N=59) | SS3: Placebo (N=385) | SS3: Upadacitinib 7.5 mg (N=20) | SS3: Upadacitinib 15 mg (N=323) | SS3: Upadacitinib 30 mg (N=316)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CATARACT (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANAL FISTULA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COLITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COLITIS ULCERATIVE (Gastrointestinal disorders) | 2 (3) | 0 (0) | 1 (1) | 4 (5) | 3 (3) | 5 (6) | 2 (2) | 1 (1) | 1 (1) | 9 (9) | 0 (0) | 1 (1) | 3 (3)
COLON DYSPLASIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIAPHRAGMATIC HERNIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ILEUS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PANCREATITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DEVICE INTOLERANCE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HEPATITIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LIVER DISORDER (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ABDOMINAL ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ACUTE ENDOCARDITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ANAL ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
APPENDICITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ARTHRITIS BACTERIAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BREAST ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BRONCHITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BURSITIS INFECTIVE (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
CELLULITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
GASTROENTERITIS NOROVIRUS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
HERPES ZOSTER MENINGITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INFECTIOUS MONONUCLEOSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INFLUENZA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LARGE INTESTINE INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MASTITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MUSCLE ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMOCYSTIS JIROVECII PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA CRYPTOCOCCAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
PNEUMONIA PNEUMOCOCCAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
POST PROCEDURAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RESPIRATORY SYNCYTIAL VIRUS INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SINUSITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TONSILLITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
UROSEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VIRAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VIRAL PHARYNGITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PULMONARY CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SKIN LACERATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
THORACIC VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CHONDROMALACIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ADENOCARCINOMA OF COLON (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
INVASIVE BREAST CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
SEBORRHOEIC KERATOSIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SMALL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ANXIETY (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
DEPRESSION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
MENTAL DISORDER (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SUICIDAL IDEATION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CYSTITIS HAEMORRHAGIC (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CERVICAL DYSPLASIA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NONINFECTIVE BRONCHITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
ERYTHEMA NODOSUM (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PANNICULITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ABORTION INDUCED (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPOTENSION (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SS1: Placebo (N=46) | SS1: Upadacitinib 7.5 mg (N=47) | SS1: Upadacitinib 15 mg (N=49) | SS1: Upadacitinib 30 mg (N=117) | SS1: Upadacitinib 45 mg (N=123) | SS2: Placebo (N=155) | SS2: Upadacitinib 45 mg (N=319) | SS2: Placebo/Upadacitinib 45 mg (N=85) | SS2: Upadacitinib 45 mg/Upadacitinib 45 mg (N=59) | SS3: Placebo (N=385) | SS3: Upadacitinib 7.5 mg (N=20) | SS3: Upadacitinib 15 mg (N=323) | SS3: Upadacitinib 30 mg (N=316)
ANAEMIA (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 3 (3) | 4 (4) | 1 (1) | 9 (9) | 8 (8) | 5 (5) | 1 (1) | 20 (24) | 1 (2) | 11 (12) | 7 (7)
LYMPHOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 6 (7) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 3 (4) | 1 (1)
CERUMEN IMPACTION (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CATARACT (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (2) | 1 (1) | 2 (2)
VISUAL IMPAIRMENT (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 5 (5)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 4 (5) | 1 (1) | 2 (2) | 8 (8) | 1 (2) | 8 (9) | 5 (5)
ABDOMINAL TENDERNESS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
APHTHOUS ULCER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 1 (1) | 4 (4)
COLITIS ULCERATIVE (Gastrointestinal disorders) | 4 (4) | 1 (1) | 2 (2) | 4 (4) | 3 (3) | 16 (16) | 1 (1) | 2 (2) | 1 (1) | 101 (110) | 3 (3) | 40 (47) | 24 (25)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 6 (6) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 4 (5) | 7 (7)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 2 (2) | 2 (2)
NAUSEA (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 8 (8) | 0 (0) | 3 (3) | 4 (5) | 1 (1) | 0 (0) | 6 (7) | 1 (1) | 6 (6) | 7 (7)
PERIANAL ERYTHEMA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
INFLUENZA LIKE ILLNESS (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
PSEUDOPOLYP (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 1 (1) | 1 (1) | 0 (0) | 5 (5) | 1 (1) | 2 (3) | 8 (8) | 6 (7) | 0 (0) | 11 (13) | 1 (1) | 10 (10) | 18 (19)
BRONCHITIS (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 4 (4) | 1 (1) | 4 (4) | 2 (2)
CYSTITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 2 (3)
EAR INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 3 (3)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 3 (3) | 0 (0) | 0 (0) | 10 (10) | 15 (16)
INFLUENZA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 4 (4) | 1 (2) | 10 (10) | 8 (10)
NASOPHARYNGITIS (Infections and infestations) | 3 (3) | 1 (1) | 3 (3) | 3 (3) | 4 (4) | 6 (6) | 15 (16) | 4 (4) | 1 (1) | 27 (28) | 0 (0) | 31 (40) | 30 (43)
ORAL HERPES (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 4 (4) | 2 (2) | 0 (0) | 7 (8) | 1 (1) | 6 (8) | 9 (11)
PULPITIS DENTAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 0 (0)
SKIN CANDIDA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 4 (4) | 3 (3) | 6 (7) | 6 (6) | 8 (9) | 0 (0) | 0 (0) | 11 (12) | 2 (2) | 19 (20) | 15 (18)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 3 (3) | 3 (3) | 2 (3) | 0 (0) | 9 (10) | 2 (2) | 10 (13) | 4 (6)
VAGINAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 2 (2) | 5 (5) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 0 (0) | 0 (0) | 3 (3) | 4 (4) | 8 (8) | 3 (3) | 16 (18) | 5 (5) | 4 (4) | 7 (7) | 0 (0) | 20 (21) | 21 (25)
HAEMOGLOBIN DECREASED (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 2 (3)
LYMPHOCYTE COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 6 (7) | 5 (6)
LYMPHOCYTE COUNT INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
DECREASED APPETITE (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (5) | 1 (1) | 3 (3) | 0 (0)
IRON DEFICIENCY (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 3 (3) | 7 (7) | 5 (5) | 0 (0) | 0 (0) | 28 (28) | 4 (5) | 19 (19) | 8 (9)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 15 (15) | 1 (1) | 11 (11) | 4 (4)
BURSITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 2 (2) | 1 (1)
OSTEOPENIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 6 (6)
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MELANOCYTIC NAEVUS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
SKIN PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
HEADACHE (Nervous system disorders) | 5 (5) | 4 (4) | 4 (4) | 9 (9) | 8 (9) | 4 (4) | 13 (16) | 4 (4) | 2 (3) | 16 (16) | 0 (0) | 10 (10) | 14 (16)
DEPRESSED MOOD (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
IRRITABILITY (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 4 (4) | 2 (2) | 5 (5) | 2 (2) | 1 (1) | 6 (6) | 2 (2) | 6 (6) | 4 (5)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 2 (2)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 4 (4) | 0 (0) | 1 (1) | 6 (6) | 1 (1) | 0 (0) | 6 (6) | 1 (1) | 5 (5) | 8 (8)
PULMONARY MASS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
ACNE (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 6 (6) | 6 (6) | 1 (1) | 15 (15) | 2 (2) | 1 (1) | 8 (8) | 0 (0) | 7 (8) | 11 (14)
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 9 (12) | 1 (1) | 2 (2) | 2 (2)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 1 (1) | 1 (1) | 8 (8) | 0 (0) | 1 (1) | 14 (14) | 2 (2) | 9 (9) | 14 (15)
ROSACEA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2021-05-10): https://cdn.clinicaltrials.gov/large-docs/35/NCT02819635/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-20): https://cdn.clinicaltrials.gov/large-docs/35/NCT02819635/SAP_001.pdf